CLINICAL TRIAL: NCT02391948
Title: Developmental Trajectories of Impairments, Health, and Participation of Children With Cerebral Palsy
Brief Title: On Track: Monitoring Development of Children With Cerebral Palsy or Gross Motor Delay
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Sarah Westcott McCoy, Professor, Rehabilitation Medicine, University of Washington
Other Study IDs: 43611
Record Dates: First submitted 2014-11-23; First posted 2015-03-18 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Gross motor delay
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The On Track Study is a large multi-site collaboration involving researchers, therapists, families, and children with cerebral palsy (CP) from across Canada and the United States. The researchers need to better understand how young children who have difficulties with movement activities progress and develop in their balance abilities, fitness, strength, health, range of motion, self-care, everyday play, and activity participation.

This study will determine how young children with cerebral palsy or gross motor delays progress in many aspects of their physical development and participation in daily life. The information collected from this study will help therapists and parents monitor if a child is developing as expected in his or her physical development and participation. Then, the health care professionals working with children can use the results of this study, in combination with the previously completed Move & PLAY study results, to provide the services that are most beneficial and meaningful for each child and their family members.

DETAILED DESCRIPTION:
Trained therapist assessors will measure the primary and secondary impairments (i.e., balance, range of motion limitations, and strength) on 5 occasions (6-months apart over 2 years). Parents will complete questionnaires to track changes in the child's endurance, health conditions, and participation in self-care and recreation activities, at the same data collection points. The researchers will use these 5 data collection points to develop reference percentiles and will present the data so that therapists can assist families to determine if children with CP are developing as expected, better than expected, or more poorly than expected, depending on their functional ability levels.

The researchers will create longitudinal developmental curves for impairments, health conditions, and participation variables by estimating the average pattern of change, important individual variations in the pattern of change between children, and the degree of consistency over time within children. Establishment of longitudinal developmental curves will provide easily understood and useful tools for families and service providers to discuss questions about how well their children are doing in relationship to other children with CP of similar functional ability levels. The researchers will then utilize service data collected from parents and children's progress on the longitudinal developmental curves to develop recommendations for rehabilitation service provision for children with CP across functional ability levels. Having this information should assist with collaborative decision-making among family members and service providers that efficiently utilizes rehabilitation services to meet families' goals.

An additional sub-study is to collect direct physical activity measurements from a sub-set of the children in the larger study. These data will be examined in relationship to other measures of endurance and participation.

ELIGIBILITY:
Inclusion Criteria:

Families with a child who has a diagnosis of cerebral palsy or delayed motor development with muscle stiffness and difficulties with balance and moving.

Certain geographical areas of Canada and the US.

Exclusion Criteria:

Children will be excluded if they have: 1) Diagnosis other than cerebral palsy (such as autism, Down syndrome, spinal cord injury, acute head injury, muscle disorder, developmental syndrome, genetic disorder); 2) Gross motor delay without associated problems with muscle tone, balance, and active movement; 3) are wards of the state; and 4) Families who do not speak English, French, or Spanish will not be eligible to participate in this study.

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cerebral palsy or gross motor delay and CP motor symptoms, ages 18 month to 12 years, and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 724 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Westcott McCoy, PhD, PT, Principal Investigator — University of Washington
Locations (5):
- United States (4):
  - Mercer University, Atlanta, Georgia
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Drexel University, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington
- University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Population: Children with cerebral palsy of gross motor delay, ages 18 month to 11 years, and their parents.
  Sampling Method: Non-Probability Sample. Participants Recruited for 2-Visit or 5-Visit Study.
Pre-assignment Details: N=724 participants agreed to participate in the study following completion of the informed consent process. The number of participants "Started" (N=708) is different from the number of participants "Enrolled" (N=724) because N=16 were Enrolled, and Not Started for the following Reasons:
  Death = 1. Lost to Follow-up = 4. Ineligible = 11.
Groups:
- Gross Motor Function Classification System (GMFCS) Level I: The GMFCS is classification system based on functional body movement ability. GMFCS levels vary from I to V, with a level closest to I reflecting higher function. The general descriptions of a child at 6 to 12 years of age are: I: Walks without limitations. Descriptors for five levels vary by the age of the child.
- Gross Motor Function Classification System (GMFCS) Level II: The GMFCS is classification system based on functional body movement ability. GMFCS levels vary from I to V, with a level closest to I reflecting higher function. The general descriptions of a child at 6 to 12 years of age are: II: Walks with limitations. Descriptors for five levels vary by the age of the child.
- Gross Motor Function Classification System (GMFCS) Level III: The GMFCS is classification system based on functional body movement ability. GMFCS levels vary from I to V, with a level closest to I reflecting higher function. The general descriptions of a child at 6 to 12 years of age are: III: Walks using a handheld mobility device. Descriptors for five levels vary by the age of the child.
- Gross Motor Function Classification System (GMFCS) Level IV: The GMFCS is classification system based on functional body movement ability. GMFCS levels vary from I to V, with a level closest to I reflecting higher function. The general descriptions of a child at 6 to 12 years of age are: IV: Self mobility with Limitations; may use powered mobility. Descriptors for five levels vary by the age of the child.
- Gross Motor Function Classification System (GMFCS) Level V: The GMFCS is classification system based on functional body movement ability. GMFCS levels vary from I to V, with a level closest to I reflecting higher function. The general descriptions of a child at 6 to 12 years of age are: V: Transported in manual wheelchair. Descriptors for five levels vary by the age of the child.
Period: Baseline
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Started | 227 | 161 | 80 | 129 | 111
Completed | 227 | 161 | 80 | 129 | 111
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 6-month Assessment
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Started | 227 | 161 | 80 | 129 | 111
Completed | 148 | 105 | 49 | 84 | 85
Not Completed | 79 | 56 | 31 | 45 | 26
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 0
Not completed — Lost to Follow-up | 4 | 5 | 2 | 3 | 1
Not completed — Medical issue/illness | 1 | 1 | 0 | 0 | 0
Not completed — Not able to schedule visit in timeframe | 6 | 8 | 4 | 5 | 0
Not completed — In 2-visit study (6-month N/A) | 68 | 42 | 24 | 35 | 24
Period: 12-month Assessment
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Started | 225 (Started at 12-month is not equal to Completed at 6-month: 77 of the Not Completed remained active.) | 156 (Started at 12-month is not equal to Completed at 6-month: 51 of the Not Completed remained active.) | 77 (Started at 12-month is not equal to Completed at 6-month: 28 of the Not Completed remained active.) | 125 (Started at 12-month is not equal to Completed at 6-month: 41 of the Not Completed remained active.) | 109 (Started at 12-month is not equal to Completed at 6-month: 24 of the Not Completed remained active.)
Completed | 217 | 147 | 73 | 116 | 103
Not Completed | 8 | 9 | 4 | 9 | 6
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 5 | 4 | 4 | 4 | 5
Not completed — Medical issue/illness | 0 | 1 | 0 | 1 | 0
Not completed — Not able to schedule visit in timeframe | 2 | 4 | 0 | 2 | 1
Period: 18-month Assessment
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Started | 219 (Started at 18-month is not equal to Completed at 12-month: 2 of the Not Completed remained active.) | 151 (Started at 18-month is not equal to Completed at 12-month: 4 of the Not Completed remained active.) | 74 (Started at 18-month is not equal to Completed at 12-month: 1 of the Not Completed remained active.) | 119 (Started at 18-month is not equal to Completed at 12-month: 3 of the Not Completed remained active.) | 105 (Started at 18-month is not equal to Completed at 12-month: 2 of the Not Completed remained active.)
Completed | 147 | 101 | 48 | 83 | 75
Not Completed | 72 | 50 | 26 | 36 | 30
Not completed — Death | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 6 | 2 | 2 | 3
Not completed — Not able to schedule visit in timeframe | 3 | 3 | 2 | 1 | 4
Not completed — In 2-visit study (18- and 24-month N/A) | 66 | 41 | 22 | 31 | 22
Period: 24-month Assessment
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Started | 149 (Started at 24-month is not equal to Completed at 18-month: 2 of the Not Completed remained active.) | 107 (Started at 24-month is not equal to Completed at 18-month: 6 of the Not Completed remained active.) | 51 (Started at 24-month is not equal to Completed at 18-month: 3 of the Not Completed remained active.) | 84 (Started at 24-month is not equal to Completed at 18-month: 1 of the Not Completed remained active.) | 79 (Started at 24-month is not equal to Completed at 18-month: 4 of the Not Completed remained active.)
Completed | 135 | 97 | 48 | 75 | 69
Not Completed | 14 | 10 | 3 | 9 | 10
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 5 | 4 | 0 | 0 | 0
Not completed — Medical issue/illness | 0 | 0 | 1 | 0 | 0
Not completed — Not able to schedule visit in timeframe | 8 | 5 | 2 | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V | Total
Number analyzed (Participants) | 227 | 161 | 80 | 129 | 111 | 708
Age, Continuous [Mean (Standard Deviation); unit: months]
  Age in Months at Baseline | 70.1 (33.5) | 75.6 (31.2) | 71.3 (31.5) | 69.6 (29.5) | 75.2 (34.3) | 72.2 (32.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 67 | 42 | 48 | 50 | 312
  Male | 122 | 94 | 38 | 81 | 61 | 396
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 15 | 4 | 11 | 6 | 49
  Not Hispanic or Latino | 214 | 142 | 76 | 117 | 105 | 654
  Unknown or Not Reported | 0 | 4 | 0 | 1 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 6 | 2 | 2 | 15
  Asian | 9 | 13 | 2 | 11 | 5 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 15 | 6 | 14 | 10 | 60
  White | 170 | 114 | 55 | 87 | 77 | 503
  More than one race | 30 | 12 | 8 | 14 | 17 | 81
  Unknown or Not Reported | 1 | 4 | 3 | 1 | 0 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 121 | 82 | 39 | 64 | 41 | 347
  United States | 106 | 79 | 41 | 65 | 70 | 361

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Assessment of Balance (ECAB)
Description: The ECAB addresses postural control and balance across the developmental sequence. Part I has 7 items (with numbers 1,4,5,6,7 scored bilaterally): 1) lateral head righting, 2) head righting in extension, 3) head righting in flexion, 4) rotation in the trunk, 5) equilibrium reactions in sitting, 6) protective extension to the side, and 7) protective extension backwards. The items are scored on a scale of 0 = no response to 3 = complete & consistent response. Part II has 6 items: 1) sitting with back unsupported but feet supported, 2) moving from sitting to standing, 3) standing unsupported with eyes closed, 4) standing unsupported with feet together, 5) turning 360 degrees in standing unsupported, 6) placing alternate foot on the step while standing unsupported. These items are scored on a variable scale, which is weighted due to the increased difficulty of the items. Part I and Part II item scores are summed for a total score between 0-100. A higher score represents better balance.
Time Frame: up to 24-months
Population: The overall N=708 available at Baseline is represented under Overall Number of Participants Analyzed. Available N at each time point is described under Participant Flow. Within each time point, there are two rows for age (under 6 years, 6 years and older).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 227 | 161 | 80 | 129 | 111
units on a scale
  Baseline: under 6 years: number analyzed (Participants) | 124 | 71 | 37 | 66 | 49
  Baseline: under 6 years | 79.4 (19.6) | 61.1 (19.2) | 38.0 (14.8) | 23.0 (8.8) | 7.3 (5.1)
  Baseline: 6 years and older: number analyzed (Participants) | 103 | 90 | 43 | 63 | 62
  Baseline: 6 years and older | 97.4 (5.1) | 86.0 (15.8) | 44.3 (14.3) | 24.7 (10.0) | 6.4 (6.8)
  6-month assessment: under 6 years: number analyzed (Participants) | 69 | 44 | 21 | 35 | 34
  6-month assessment: under 6 years | 80.4 (18.9) | 61.6 (19.8) | 37.6 (12.7) | 26.1 (8.4) | 8.1 (7.5)
  6-month assessment: 6 years and older: number analyzed (Participants) | 79 | 61 | 28 | 49 | 51
  6-month assessment: 6 years and older | 97.4 (5.2) | 86.1 (16.9) | 49.0 (17.0) | 24.8 (11.9) | 7.2 (6.6)
  12-month assessment: under 6 years: number analyzed (Participants) | 93 | 49 | 26 | 46 | 41
  12-month assessment: under 6 years | 86.3 (14.3) | 64.9 (20.8) | 37.5 (7.9) | 26.3 (7.9) | 7.6 (6.3)
  12-month assessment: 6 years and older: number analyzed (Participants) | 124 | 98 | 47 | 70 | 62
  12-month assessment: 6 years and older | 98.1 (4.4) | 86.9 (15.8) | 50.6 (19.0) | 25.0 (10.9) | 8.0 (7.9)
  18-month assessment: under 6 years: number analyzed (Participants) | 58 | 34 | 17 | 26 | 24
  18-month assessment: under 6 years | 86.6 (15.1) | 62.8 (18.9) | 41.4 (12.3) | 29.3 (8.2) | 7.7 (7.1)
  18-month assessment: 6 years and older: number analyzed (Participants) | 89 | 67 | 31 | 57 | 51
  18-month assessment: 6 years and older | 97.9 (4.8) | 86.9 (16.5) | 52.6 (19.9) | 25.9 (11.7) | 7.4 (6.9)
  24-month assessment: under 6 years: number analyzed (Participants) | 46 | 24 | 17 | 18 | 18
  24-month assessment: under 6 years | 89.8 (14.5) | 62.2 (17.8) | 40.7 (11.6) | 28.5 (8.0) | 7.1 (6.2)
  24-month assessment: 6 years and older: number analyzed (Participants) | 89 | 73 | 31 | 57 | 51
  24-month assessment: 6 years and older | 98.4 (3.7) | 87.0 (16.1) | 54.3 (21.9) | 24.9 (10.9) | 7.1 (6.1)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; Test type: Other; mean population value age 12 = 98.3, 95% CI 2-sided [97.8 to 98.6]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; Test type: Other; mean population value age 12 = 89.1, 95% CI 2-sided [86.6 to 91.1]
Statistical Analysis 3: Comparison: Gross Motor Function Classification System (GMFCS) Level III; Test type: Other; mean population value age 12 = 50.1, 95% CI 2-sided [46.5 to 53.6]
Statistical Analysis 4: Comparison: Gross Motor Function Classification System (GMFCS) Level IV; Test type: Other; mean population value age 12 = 25.3, 95% CI 2-sided [23.7 to 27.0]
Statistical Analysis 5: Comparison: Gross Motor Function Classification System (GMFCS) Level V; Test type: Other; mean population value age 12 = 6.48, 95% CI 2-sided [5.66 to 7.38]

2. Primary Outcome: Spinal Alignment and Range of Motion Measure (SAROMM)
Description: The SAROMM addresses joint range of motion, extensibility, and spinal alignment. The Spinal Alignment Subscale contains 4 items and the Range of Motion and Extensibility Subscale has 22 items. Each item is scored on a 5-point Likert scale, with 0 = normal alignment and range with active correction, 1 = normal alignment and range with passive correction, and 2, 3, and 4 indicating fixed deformities or contractures that are "mild", "moderate", or "severe" based on pre-specified cut points, and supported by photographs in the training manual. Scores are reported by calculating the average of scores across all 26 items. Scores range from 0-4. A lower score represents better range of motion and alignment.
Time Frame: up to 24-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 227 | 161 | 80 | 129 | 111
units on a scale
  Baseline: under 6 years: number analyzed (Participants) | 124 | 71 | 37 | 66 | 49
  Baseline: under 6 years | 0.3 (0.3) | 0.6 (0.4) | 0.9 (0.4) | 1.1 (0.5) | 1.4 (0.5)
  Baseline: 6 years and older: number analyzed (Participants) | 103 | 90 | 43 | 63 | 62
  Baseline: 6 years and older | 0.4 (0.3) | 0.6 (0.4) | 1.0 (0.5) | 1.5 (0.6) | 1.9 (0.6)
  6-month assessment: under 6 years: number analyzed (Participants) | 69 | 44 | 21 | 35 | 34
  6-month assessment: under 6 years | 0.3 (0.3) | 0.6 (0.4) | 0.8 (0.3) | 1.0 (0.6) | 1.2 (0.6)
  6-month assessment: 6 years and older: number analyzed (Participants) | 79 | 61 | 28 | 49 | 51
  6-month assessment: 6 years and older | 0.4 (0.3) | 0.6 (0.4) | 0.8 (0.4) | 1.3 (0.6) | 1.9 (0.6)
  12-month assessment: under 6 years: number analyzed (Participants) | 93 | 49 | 26 | 46 | 41
  12-month assessment: under 6 years | 0.3 (0.2) | 0.6 (0.4) | 0.8 (0.4) | 1.1 (0.5) | 1.4 (0.6)
  12-month assessment: 6 years and older: number analyzed (Participants) | 124 | 98 | 47 | 70 | 62
  12-month assessment: 6 years and older | 0.4 (0.3) | 0.6 (0.4) | 0.9 (0.4) | 1.3 (0.5) | 2.0 (0.6)
  18-month assessment: under 6 years: number analyzed (Participants) | 58 | 34 | 17 | 26 | 24
  18-month assessment: under 6 years | 0.3 (0.3) | 0.6 (0.4) | 0.8 (0.4) | 1.0 (0.5) | 1.3 (0.6)
  18-month assessment: 6 years and older: number analyzed (Participants) | 89 | 67 | 31 | 57 | 51
  18-month assessment: 6 years and older | 0.4 (0.3) | 0.7 (0.4) | 0.9 (0.3) | 1.3 (0.6) | 1.9 (0.6)
  24-month assessment: under 6 years: number analyzed (Participants) | 46 | 24 | 17 | 18 | 18
  24-month assessment: under 6 years | 0.4 (0.3) | 0.7 (0.4) | 0.8 (0.5) | 1.0 (0.6) | 1.4 (0.7)
  24-month assessment: 6 years and older: number analyzed (Participants) | 89 | 73 | 31 | 57 | 51
  24-month assessment: 6 years and older | 0.4 (0.3) | 0.6 (0.4) | 0.9 (0.5) | 1.3 (0.6) | 2.0 (0.6)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; Test type: Other; mean population value age 12 = 0.44, 95% CI 2-sided [0.38 to 0.49]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; Test type: Other; mean population value age 12 = 0.68, 95% CI 2-sided [0.60 to 0.77]
Statistical Analysis 3: Comparison: Gross Motor Function Classification System (GMFCS) Level III; Test type: Other; mean population value age 12 = 0.93, 95% CI 2-sided [0.79 to 1.07]
Statistical Analysis 4: Comparison: Gross Motor Function Classification System (GMFCS) Level IV; Test type: Other; mean population value age 12 = 1.38, 95% CI 2-sided [1.22 to 1.54]
Statistical Analysis 5: Comparison: Gross Motor Function Classification System (GMFCS) Level V; Test type: Other; mean population value age 12 = 2.16, 95% CI 2-sided [2.01 to 2.31]

3. Primary Outcome: Functional Strength Assessment (FSA)
Description: The FSA addresses force production ability in the neck and trunk flexor and extensor and bilateral hip and knee extensor and shoulder flexor muscle groups. Each muscle group is rated on a five-point ordinal scale from 1 = only flicker of contraction or just initiates movement against gravity to 5 = full available range against gravity and strong resistance. Scores are reported by calculating the average of scores across all 8 items. Scores range from 1 to 5. A higher score represents better force production ability.
Time Frame: up to 24-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 227 | 161 | 80 | 129 | 111
units on a scale
  Baseline: under 6 years: number analyzed (Participants) | 124 | 71 | 37 | 66 | 49
  Baseline: under 6 years | 4.0 (0.7) | 3.6 (0.6) | 3.1 (0.6) | 2.6 (0.7) | 1.8 (0.7)
  Baseline: 6 years and older: number analyzed (Participants) | 103 | 90 | 43 | 63 | 62
  Baseline: 6 years and older | 4.5 (0.5) | 4.1 (0.6) | 3.6 (0.8) | 2.7 (0.8) | 1.5 (0.5)
  6-month assessment: under 6 years: number analyzed (Participants) | 69 | 44 | 21 | 35 | 34
  6-month assessment: under 6 years | 4.0 (0.7) | 3.6 (0.6) | 3.1 (0.6) | 2.7 (0.6) | 1.7 (0.6)
  6-month assessment: 6 years and older: number analyzed (Participants) | 79 | 61 | 28 | 49 | 51
  6-month assessment: 6 years and older | 4.5 (0.5) | 4.1 (0.6) | 3.6 (0.8) | 2.7 (0.8) | 1.6 (0.6)
  12-month assessment: under 6 years: number analyzed (Participants) | 93 | 49 | 26 | 46 | 41
  12-month assessment: under 6 years | 4.2 (0.6) | 3.7 (0.6) | 3.2 (0.7) | 2.8 (0.5) | 1.8 (0.7)
  12-month assessment: 6 years and older: number analyzed (Participants) | 124 | 98 | 47 | 70 | 62
  12-month assessment: 6 years and older | 4.6 (0.4) | 4.2 (0.6) | 3.6 (0.8) | 2.7 (0.8) | 1.6 (0.5)
  18-month assessment: under 6 years: number analyzed (Participants) | 58 | 34 | 17 | 26 | 24
  18-month assessment: under 6 years | 4.0 (0.7) | 3.5 (0.7) | 3.1 (0.7) | 2.9 (0.6) | 1.7 (0.6)
  18-month assessment: 6 years and older: number analyzed (Participants) | 89 | 67 | 31 | 57 | 51
  18-month assessment: 6 years and older | 4.5 (0.5) | 4.1 (0.7) | 3.7 (0.7) | 2.8 (0.8) | 1.7 (0.5)
  24-month assessment: under 6 years: number analyzed (Participants) | 46 | 24 | 17 | 18 | 18
  24-month assessment: under 6 years | 4.1 (0.6) | 3.6 (0.8) | 3.1 (0.6) | 2.7 (0.7) | 1.5 (0.5)
  24-month assessment: 6 years and older: number analyzed (Participants) | 89 | 73 | 31 | 57 | 51
  24-month assessment: 6 years and older | 4.6 (0.4) | 4.1 (0.7) | 3.8 (0.8) | 2.9 (0.9) | 1.6 (0.5)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; Test type: Other; mean population value = 4.49, 95% CI 2-sided [4.43 to 4.54]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; Test type: Other; mean population value = 4.10, 95% CI 2-sided [3.99 to 4.20]
Statistical Analysis 3: Comparison: Gross Motor Function Classification System (GMFCS) Level III; Test type: Other; mean population value = 3.99, 95% CI 2-sided [3.75 to 4.25]
Statistical Analysis 4: Comparison: Gross Motor Function Classification System (GMFCS) Level IV; Test type: Other; mean population value = 2.95, 95% CI 2-sided [2.73 to 3.19]
Statistical Analysis 5: Comparison: Gross Motor Function Classification System (GMFCS) Level V; Test type: Other; mean population value = 1.59, 95% CI 2-sided [1.44 to 1.75]

4. Primary Outcome: Six and One-minute Walk Test (6MWT, 1MWT)
Description: The 6MWT and 1MWT are submaximal, clinical exercise tests, in which the total distance traveled in 1-minute and 6-minutes, under controlled conditions, are measured. Within this study, the 6MWT/1MWT was conducted indoors or outdoors on a large, flat, hard terrain for children who were 3 years or older and who were walking without another person's assistance (GMFCS I, II, III). A surveyor's measure wheel was used to calculate the total distance (# of feet) walked and a stopwatch to keep track of the allocated time. Standardized directions are used to encourage the child to walk as far as possible in the time.
Time Frame: up to 24-months
Population: The available N for 6MWT at 12M (highest #) is represented under Overall # Analyzed. For each time point, there are 2 rows for age. Of the available N at each time point (see Participant Flow), the Walk Test was given only to GMFCS Level I, II, or III age 3yrs+. The 1MWT was given to a smaller subset of children in the Physical Activity Sub-Study.
Measure: Mean (Standard Deviation); unit: Feet
Groups:
- Gross Motor Function Classification System (GMFCS) Level II; Gross Motor Function Classification System (GMFCS) Level III: The GMFCS is classification system based on functional body movement ability. GMFCS levels vary from I to V, with a level closest to I reflecting higher function. The general descriptions of a child at 6 to 12 years of age are: I: Walks without limitations. Descriptors for five levels vary by the age of the child.
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III
Number analyzed (Participants) | 201 | 144 | 63
Feet
  6MWT, Baseline: under 6 years: number analyzed (Participants) | 73 | 48 | 20
  6MWT, Baseline: under 6 years | 1080.3 (273.6) | 697.3 (347.1) | 396.2 (317.6)
  6MWT, Baseline: 6 years and older: number analyzed (Participants) | 103 | 90 | 42
  6MWT, Baseline: 6 years and older | 1386.2 (342.5) | 1041.8 (303.4) | 616.9 (307.0)
  6MWT, 6-month assessment: under 6 years: number analyzed (Participants) | 52 | 33 | 9
  6MWT, 6-month assessment: under 6 years | 1012.8 (301.6) | 611.1 (314.5) | 359.5 (273.8)
  6MWT, 6-month assessment: 6 years and older: number analyzed (Participants) | 79 | 61 | 27
  6MWT, 6-month assessment: 6 years and older | 1370.0 (321.1) | 1075.0 (322.1) | 574.0 (312.9)
  6MWT, 12-month assessment: under 6 years: number analyzed (Participants) | 77 | 46 | 18
  6MWT, 12-month assessment: under 6 years | 1026.7 (282.7) | 658.9 (339.4) | 314.6 (237.1)
  6MWT, 12-month assessment: 6 years and older: number analyzed (Participants) | 124 | 98 | 45
  6MWT, 12-month assessment: 6 years and older | 1378.4 (325.3) | 1047.7 (356.5) | 690.7 (261.1)
  6MWT, 18-month assessment: under 6 years: number analyzed (Participants) | 57 | 34 | 15
  6MWT, 18-month assessment: under 6 years | 1020.1 (311.5) | 601.6 (239.0) | 331.6 (218.2)
  6MWT, 18-month assessment: 6 years and older: number analyzed (Participants) | 89 | 67 | 30
  6MWT, 18-month assessment: 6 years and older | 1351.1 (324.4) | 1109.0 (324.2) | 636.5 (312.9)
  6MWT, 24-month assessment: under 6 years: number analyzed (Participants) | 46 | 24 | 13
  6MWT, 24-month assessment: under 6 years | 1197.6 (1178.3) | 613.0 (239.8) | 413.8 (226.0)
  6MWT, 24-month assessment: 6 years and older: number analyzed (Participants) | 89 | 73 | 29
  6MWT, 24-month assessment: 6 years and older | 1401.7 (288.6) | 1113.7 (336.6) | 616.4 (319.3)
  1MWT, Baseline: under 6 years: number analyzed (Participants) | 0 | 3 | 1
  1MWT, Baseline: under 6 years |  | 118.93 (79.28) | 15.30 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  1MWT, Baseline: 6 years and older: number analyzed (Participants) | 5 | 5 | 2
  1MWT, Baseline: 6 years and older | 263.18 (49.23) | 120.13 (74.74) | 78.42 (13.31)
  1MWT, 6-month assessment: under 6 years: number analyzed (Participants) | 4 | 4 | 1
  1MWT, 6-month assessment: under 6 years | 201.28 (7.64) | 128.65 (33.22) | 28.40 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  1MWT, 6-month assessment: 6 years and older: number analyzed (Participants) | 11 | 6 | 3
  1MWT, 6-month assessment: 6 years and older | 239.40 (68.41) | 234.12 (63.15) | 121.60 (28.76)
  1MWT, 12-month assessment: under 6 years: number analyzed (Participants) | 4 | 3 | 2
  1MWT, 12-month assessment: under 6 years | 215.37 (28.96) | 150.58 (56.83) | 70.95 (4.60)
  1MWT, 12-month assessment: 6 years and older: number analyzed (Participants) | 15 | 11 | 5
  1MWT, 12-month assessment: 6 years and older | 242.51 (66.46) | 211.11 (67.26) | 102.62 (32.93)
  1MWT, 18-month assessment: under 6 years: number analyzed (Participants) | 3 | 1 | 1
  1MWT, 18-month assessment: under 6 years | 190.40 (7.81) | 107.00 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 89.10 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  1MWT, 18-month assessment: 6 years and older: number analyzed (Participants) | 14 | 10 | 5
  1MWT, 18-month assessment: 6 years and older | 242.18 (57.16) | 208.03 (44.36) | 103.38 (49.29)
  1MWT, 24-month assessment: under 6 years: number analyzed (Participants) | 1 | 0 | 1
  1MWT, 24-month assessment: under 6 years | 194.00 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |  | 77.40 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  1MWT, 24-month assessment: 6 years and older: number analyzed (Participants) | 14 | 15 | 5
  1MWT, 24-month assessment: 6 years and older | 254.34 (56.63) | 239.30 (157.77) | 84.34 (44.86)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; Test type: Other; mean population value = 1362.3, 95% CI 2-sided [1313.6 to 1410.7]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; Test type: Other; mean population value = 1096.33, 95% CI 2-sided [1028.80 to 1158.62]
Statistical Analysis 3: Comparison: Gross Motor Function Classification System (GMFCS) Level III; Test type: Other; mean population value = 592.62, 95% CI 2-sided [533.79 to 652.72]

5. Primary Outcome: Early Activity Scale for Endurance (EASE)
Description: The EASE includes 4 activity-based items requiring parents to rate their children's levels of energy, the frequency and need for rest, and the average amount of time their children can engage in physical activity. Scoring for each item is on a Likert scale of 1-5 with the value of 1 = "Never" to 5 = "Always". The four questions include: 1) "my child's physical activity level is similar to other children his or her age," 2) "my child has a high physical energy level and rarely needs to take rests when moving himself or herself around during daily activities and play time," 3) "my child does enough activity so that he or she is breathing quickly or gets flushing in his or her face at least one time each day," and 4) "my child spends a lot of his or her play or free time doing activities that require lots of physical energy." Scores are reported by calculating the average across all 4 questions. Scores range from 1 to 5. A higher score represents better endurance for activity.
Time Frame: up to 24-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 227 | 161 | 80 | 129 | 111
units on a scale
  Baseline: under 6 years: number analyzed (Participants) | 124 | 71 | 37 | 66 | 49
  Baseline: under 6 years | 4.0 (0.7) | 3.6 (0.8) | 3.3 (0.7) | 2.7 (0.9) | 1.9 (1.0)
  Baseline: 6 years and older: number analyzed (Participants) | 103 | 90 | 43 | 63 | 62
  Baseline: 6 years and older | 3.7 (0.7) | 3.2 (0.8) | 3.0 (0.8) | 2.8 (0.9) | 1.7 (0.7)
  6-month assessment: under 6 years: number analyzed (Participants) | 69 | 44 | 21 | 35 | 34
  6-month assessment: under 6 years | 4.0 (0.7) | 3.6 (0.8) | 3.3 (0.8) | 2.8 (0.9) | 1.9 (0.9)
  6-month assessment: 6 years and older: number analyzed (Participants) | 79 | 61 | 28 | 49 | 51
  6-month assessment: 6 years and older | 3.8 (0.8) | 3.2 (0.9) | 3.1 (0.8) | 2.8 (1.0) | 1.7 (0.7)
  12-month assessment: under 6 years: number analyzed (Participants) | 93 | 49 | 26 | 46 | 41
  12-month assessment: under 6 years | 4.1 (0.6) | 3.7 (0.7) | 3.5 (0.9) | 2.7 (1.0) | 2.1 (0.9)
  12-month assessment: 6 years and older: number analyzed (Participants) | 124 | 98 | 47 | 70 | 62
  12-month assessment: 6 years and older | 3.8 (0.8) | 3.4 (0.9) | 3.2 (0.8) | 2.8 (0.9) | 1.7 (0.7)
  18-month assessment: under 6 years: number analyzed (Participants) | 58 | 34 | 17 | 26 | 24
  18-month assessment: under 6 years | 4.3 (0.7) | 3.7 (0.8) | 3.4 (0.8) | 2.6 (0.9) | 1.7 (0.7)
  18-month assessment: 6 years and older: number analyzed (Participants) | 89 | 67 | 31 | 57 | 51
  18-month assessment: 6 years and older | 3.8 (0.9) | 3.3 (1.0) | 3.1 (0.9) | 2.8 (0.9) | 1.7 (0.8)
  24-month assessment: under 6 years: number analyzed (Participants) | 46 | 24 | 17 | 18 | 18
  24-month assessment: under 6 years | 4.1 (0.7) | 3.7 (0.8) | 3.5 (0.8) | 2.9 (0.8) | 1.8 (0.7)
  24-month assessment: 6 years and older: number analyzed (Participants) | 89 | 73 | 31 | 57 | 51
  24-month assessment: 6 years and older | 3.9 (0.8) | 3.3 (0.9) | 3.1 (0.9) | 2.7 (0.9) | 1.8 (0.8)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; Test type: Other; mean population value = 3.99, 95% CI 2-sided [3.91 to 4.07]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; Test type: Other; mean population value = 3.49, 95% CI 2-sided [3.39 to 3.60]
Statistical Analysis 3: Comparison: Gross Motor Function Classification System (GMFCS) Level III; Test type: Other; mean population value = 3.23, 95% CI 2-sided [3.08 to 3.37]
Statistical Analysis 4: Comparison: Gross Motor Function Classification System (GMFCS) Level IV; Test type: Other; mean population value = 2.80, 95% CI 2-sided [2.67 to 2.93]
Statistical Analysis 5: Comparison: Gross Motor Function Classification System (GMFCS) Level V; Test type: Other; mean population value = 1.79, 95% CI 2-sided [1.67 to 1.91]

6. Primary Outcome: Child Health Conditions Questionnaire
Description: The Child Health Conditions questionnaire is a caregiver-completed measure of the extent to which health problems influence children's activities. Parents respond "yes" or "no" as to whether the child has each of the 16 health problems listed. If the child does not have a problem, a score of 0 is imputed for the next part of the question. If the child has a problem, parents are asked to judge the extent to which the problem affects the child's daily activities. This is measured using an 8-point ordinal scale from 0="does not have the problem", 1= "not at all" to 7 = "to a very great extent". Scores reported are the Child Health Conditions Impact average scores calculated by averaging across all 16 items. Scores range form 0 to 7. A higher score represents a greater impact of health conditions on daily activities.
Time Frame: up to 24-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 227 | 161 | 80 | 129 | 111
units on a scale
  Baseline: under 6 years: number analyzed (Participants) | 124 | 71 | 37 | 66 | 49
  Baseline: under 6 years | 0.5 (0.6) | 0.9 (0.7) | 0.9 (0.7) | 1.4 (0.8) | 2.1 (1.0)
  Baseline: 6 years and older: number analyzed (Participants) | 103 | 90 | 43 | 63 | 62
  Baseline: 6 years and older | 0.7 (0.6) | 1.1 (0.9) | 0.9 (0.6) | 1.5 (1.0) | 2.4 (1.1)
  6-month assessment: under 6 years: number analyzed (Participants) | 69 | 44 | 21 | 35 | 34
  6-month assessment: under 6 years | 0.5 (0.6) | 0.8 (0.6) | 0.9 (0.7) | 1.3 (0.9) | 2.2 (0.8)
  6-month assessment: 6 years and older: number analyzed (Participants) | 79 | 61 | 28 | 49 | 51
  6-month assessment: 6 years and older | 0.7 (0.7) | 1.2 (0.9) | 0.9 (0.6) | 1.4 (0.9) | 2.4 (1.1)
  12-month assessment: under 6 years: number analyzed (Participants) | 93 | 49 | 26 | 46 | 41
  12-month assessment: under 6 years | 0.4 (0.5) | 0.7 (0.6) | 0.8 (0.7) | 1.3 (0.9) | 2.2 (0.9)
  12-month assessment: 6 years and older: number analyzed (Participants) | 124 | 98 | 47 | 70 | 62
  12-month assessment: 6 years and older | 0.7 (0.7) | 1.0 (0.9) | 0.8 (0.6) | 1.5 (0.9) | 2.3 (1.1)
  18-month assessment: under 6 years: number analyzed (Participants) | 58 | 34 | 17 | 26 | 24
  18-month assessment: under 6 years | 0.5 (0.6) | 0.9 (0.8) | 1.0 (0.8) | 1.3 (0.9) | 2.2 (0.8)
  18-month assessment: 6 years and older: number analyzed (Participants) | 89 | 67 | 31 | 57 | 51
  18-month assessment: 6 years and older | 0.7 (0.6) | 1.0 (0.8) | 0.9 (0.7) | 1.3 (0.8) | 2.3 (1.0)
  24-month assessment: under 6 years: number analyzed (Participants) | 46 | 24 | 17 | 18 | 18
  24-month assessment: under 6 years | 0.6 (0.8) | 0.8 (0.6) | 0.8 (0.6) | 1.2 (1.0) | 2.4 (1.1)
  24-month assessment: 6 years and older: number analyzed (Participants) | 89 | 73 | 31 | 57 | 51
  24-month assessment: 6 years and older | 0.6 (0.6) | 1.0 (0.9) | 0.8 (0.7) | 1.4 (0.9) | 2.4 (1.0)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; Test type: Other; mean population value = 0.59, 9% CI 2-sided [0.47 to 0.72]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; Test type: Other; mean population value = 1.10, 95% CI 2-sided [0.91 to 1.30]
Statistical Analysis 3: Comparison: Gross Motor Function Classification System (GMFCS) Level III; Test type: Other; mean population value = 0.68, 95% CI 2-sided [0.48 to 0.89]
Statistical Analysis 4: Comparison: Gross Motor Function Classification System (GMFCS) Level IV; Test type: Other; mean population value = 1.38, 95% CI 2-sided [1.12 to 1.65]
Statistical Analysis 5: Comparison: Gross Motor Function Classification System (GMFCS) Level V; Test type: Other; mean population value = 2.33, 95% CI 2-sided [2.08 to 2.60]

7. Primary Outcome: Child Engagement in Daily Life Measure (CEDL): Part 1 - Participation
Description: CEDL is a 40-item caregiver-completed questionnaire to estimate children's participation. Part 1 captures participation of the child in family/community and leisure/recreational activities. Part 1 is scored on two 5-point Likert scales: 1) how often a child participates (1=almost never to 4=very often), and 2) the degree of enjoyment (1=not at all to 5 a great deal). A Rasch analysis has converted scores into 0-100 scaled scores. A higher score represents a higher degree of 'leisure.'
Time Frame: up to 24-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 227 | 161 | 80 | 129 | 111
units on a scale
  Participation, Baseline: <6yrs: number analyzed (Participants) | 124 | 71 | 37 | 66 | 49
  Participation, Baseline: <6yrs | 67.0 (13.4) | 65.1 (12.4) | 62.3 (12.6) | 55.8 (10.5) | 54.0 (12.5)
  Participation, Baseline 6yrs+: number analyzed (Participants) | 103 | 90 | 43 | 63 | 62
  Participation, Baseline 6yrs+ | 70.2 (15.4) | 63.9 (12.7) | 62.6 (10.9) | 58.9 (12.9) | 52.4 (9.7)
  Participation, 6-month assessment:<6yrs: number analyzed (Participants) | 69 | 44 | 21 | 35 | 34
  Participation, 6-month assessment:<6yrs | 67.9 (13.6) | 67.7 (12.6) | 57.8 (8.8) | 57.3 (9.3) | 53.9 (17.1)
  Participation, 6-month assessment 6yrs+: number analyzed (Participants) | 79 | 61 | 28 | 49 | 51
  Participation, 6-month assessment 6yrs+ | 70.0 (15.5) | 61.4 (12.9) | 63.0 (12.6) | 60.2 (12.4) | 50.0 (9.8)
  Participation, 12-month assessment: <6yrs: number analyzed (Participants) | 93 | 49 | 26 | 46 | 41
  Participation, 12-month assessment: <6yrs | 70.3 (13.3) | 64.2 (12.6) | 62.3 (9.7) | 56.1 (9.9) | 52.1 (9.8)
  Participation, 12-month assessment: 6yrs+: number analyzed (Participants) | 124 | 98 | 47 | 70 | 62
  Participation, 12-month assessment: 6yrs+ | 70.3 (14.1) | 64.1 (13.1) | 62.1 (12.5) | 58.1 (10.8) | 50.5 (9.9)
  Participation, 18-month assessment: <6yrs: number analyzed (Participants) | 58 | 34 | 17 | 26 | 24
  Participation, 18-month assessment: <6yrs | 69.7 (12.5) | 66.5 (14.2) | 65.4 (10.5) | 58.6 (10.2) | 54.0 (14.1)
  Participation, 18-month assessment 6yrs+: number analyzed (Participants) | 89 | 67 | 31 | 57 | 51
  Participation, 18-month assessment 6yrs+ | 69.3 (13.7) | 64.8 (14.2) | 58.3 (9.2) | 58.0 (11.2) | 48.4 (11.2)
  Participation, 24-month assessment: <6yrs: number analyzed (Participants) | 46 | 24 | 17 | 18 | 18
  Participation, 24-month assessment: <6yrs | 71.1 (16.2) | 70.7 (14.6) | 67.1 (14.2) | 56.6 (9.5) | 51.8 (14.0)
  Participation, 24-month assessment: 6yrs+: number analyzed (Participants) | 89 | 73 | 31 | 57 | 51
  Participation, 24-month assessment: 6yrs+ | 70.4 (15.3) | 65.5 (13.6) | 60.2 (12.0) | 56.3 (10.1) | 48.5 (13.7)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; Test type: Other; mean population value age 12 = 70.6, 95% CI 2-sided [69.1 to 72.0]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; Test type: Other; mean population value age 12 = 62.1, 95% CI 2-sided [59.4 to 65.0]
Statistical Analysis 3: Comparison: Gross Motor Function Classification System (GMFCS) Level III; Test type: Other; mean population value age 12 = 62.9, 95% CI 2-sided [60.9 to 65.0]
Statistical Analysis 4: Comparison: Gross Motor Function Classification System (GMFCS) Level IV; Test type: Other; mean population value age 12 = 58.2, 95% CI 2-sided [56.7 to 59.7]
Statistical Analysis 5: Comparison: Gross Motor Function Classification System (GMFCS) Level V; Test type: Other; mean population value age 12 = 51.9, 95% CI 2-sided [50.2 to 53.6]

8. Primary Outcome: Child Engagement in Daily Life Measure (CEDL): Part 2 - Self-Care
Description: CEDL is a 40-item caregiver-completed questionnaire to estimate children's participation. Part 2 measures self-care, defined as the degree that the child participates in daily feeding, dressing, bathing, and toileting. Part 2 is scored on a 5-point Likert scale from 1= 'does not do the activity' to 5= 'does the activity independently most of the time'. The scale distinguishes the need for physical assistance from a person, the ability to complete the activity under various conditions, and the amount of the activity able to complete. A Rasch analysis has converted scores into 0-100 scaled scores for both parts. A higher score represents a higher degree of self-care (Part 2) participation.
Time Frame: up to 24-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 227 | 161 | 80 | 129 | 111
units on a scale
  Self-care, Baseline: <6yrs: number analyzed (Participants) | 124 | 71 | 37 | 66 | 49
  Self-care, Baseline: <6yrs | 54.4 (12.5) | 49.0 (9.7) | 44.4 (10.0) | 33.6 (14.6) | 16.1 (12.3)
  Self-care, Baseline: 6yrs+: number analyzed (Participants) | 103 | 90 | 43 | 63 | 62
  Self-care, Baseline: 6yrs+ | 73.0 (14.4) | 62.1 (13.5) | 55.3 (9.3) | 35.8 (15.5) | 13.6 (15.1)
  Self-care, 6-month assessment: <6yrs: number analyzed (Participants) | 69 | 44 | 21 | 35 | 34
  Self-care, 6-month assessment: <6yrs | 56.3 (11.4) | 50.6 (8.8) | 44.0 (8.8) | 34.0 (14.5) | 15.6 (13.6)
  Self-care, 6-month assessment: 6yrs+: number analyzed (Participants) | 79 | 61 | 28 | 49 | 51
  Self-care, 6-month assessment: 6yrs+ | 72.1 (12.7) | 63.7 (15.8) | 56.0 (10.9) | 37.6 (16.1) | 12.1 (14.8)
  Self-care, 12-month assessment: <6yrs: number analyzed (Participants) | 93 | 49 | 26 | 46 | 41
  Self-care, 12-month assessment: <6yrs | 61.8 (12.7) | 54.0 (10.5) | 47.1 (8.2) | 37.3 (11.8) | 16.5 (13.4)
  Self-care, 12-month assessment: 6yrs+: number analyzed (Participants) | 124 | 98 | 47 | 70 | 62
  Self-care, 12-month assessment: 6yrs+ | 76.3 (14.8) | 64.5 (14.9) | 59.2 (13.4) | 36.9 (17.6) | 13.1 (16.1)
  Self-care, 18-month assessment: <6yrs: number analyzed (Participants) | 58 | 34 | 17 | 26 | 24
  Self-care, 18-month assessment: <6yrs | 61.4 (14.0) | 50.7 (12.6) | 46.7 (7.2) | 38.0 (14.4) | 18.1 (13.6)
  Self-care, 18-month assessment: 6yrs+: number analyzed (Participants) | 89 | 67 | 31 | 57 | 51
  Self-care, 18-month assessment: 6yrs+ | 75.2 (15.1) | 65.9 (16.8) | 59.3 (13.1) | 37.1 (18.2) | 13.6 (15.4)
  Self-care, 24-month assessment: <6yrs: number analyzed (Participants) | 46 | 24 | 17 | 18 | 18
  Self-care, 24-month assessment: <6yrs | 62.3 (12.8) | 53.5 (9.7) | 48.3 (6.7) | 34.6 (16.8) | 15.9 (13.8)
  Self-care, 24-month assessment: 6yrs+: number analyzed (Participants) | 89 | 73 | 31 | 57 | 51
  Self-care, 24-month assessment: 6yrs+ | 76.8 (14.4) | 66.1 (16.5) | 61.1 (15.0) | 37.5 (16.3) | 11.6 (14.0)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; Test type: Other; mean population value age 12 = 78.3, 95% CI 2-sided [76.0 to 80.4]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; Test type: Other; mean population value age 12 = 66.1, 95% CI 2-sided [63.5 to 68.5]
Statistical Analysis 3: Comparison: Gross Motor Function Classification System (GMFCS) Level III; Test type: Other; mean population value age 12; mean population value age 12 = 60.5, 95% CI 2-sided [57.3 to 63.3]
Statistical Analysis 4: Comparison: Gross Motor Function Classification System (GMFCS) Level IV; Test type: Other; mean population value age 12 = 37.9, 95% CI 2-sided [35.6 to 40.3]
Statistical Analysis 5: Comparison: Gross Motor Function Classification System (GMFCS) Level V; Test type: Other; mean population value age 12 = 14.5, 95% CI 2-sided [12.4 to 16.5]

9. Primary Outcome: Services Questionnaire
Description: The Services questionnaire is a caregiver-completed measure of the medical and rehabilitation services provided to the child in the period since the last data collection point. The variables used for the analysis of the relationship between services and four outcomes are reported. These data are: mean amount of physical, occupational, and speech and language therapy service sessions per year (recorded in 5 ordinal intensity times/year categories: 1=0-1, 2=2-30, 3=31-52, 4=53-155, 5=>156), mean family centeredness across 14 items (scored in 5 ordinal categories: 1=not at all, 2=small, 3=moderate, 4=great, 5=very great extent), mean rating of parents' perceptions that services were meeting their children's needs (scored on ordinal scale 1=not at all, 2=small, 3=moderate, 4=great extent, 5=completely), mean rating of the extent to which therapy was focused into 8 categories (scored in same ordinal categories as family centeredness above). Higher scores indicate a great amount or extent.
Time Frame: up to 24-months
Population: The overall N=708 available at Baseline is represented under Overall Number of Participants Analyzed. Available N at each time point is described under Participant Flow.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 227 | 161 | 80 | 129 | 111
units on a scale
  Intensity of services: PT Baseline | 2.2 (0.8) | 2.5 (1.0) | 2.8 (0.9) | 2.9 (1.0) | 2.9 (1.0)
  Intensity of services: PT 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Intensity of services: PT 6M | 2.2 (0.9) | 2.8 (1.0) | 3.3 (1.0) | 3.2 (1.0) | 3.2 (1.0)
  Intensity of services: PT 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Intensity of services: PT 12M | 2.0 (0.9) | 2.6 (1.1) | 3.0 (1.0) | 3.0 (1.0) | 2.9 (1.1)
  Intensity of services: PT 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Intensity of services: PT 18M | 2.1 (1.1) | 2.7 (1.2) | 3.0 (1.1) | 3.2 (1.0) | 3.1 (1.0)
  Intensity of services: PT 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Intensity of services: PT 24M | 2.0 (1.0) | 2.8 (1.1) | 3.0 (1.1) | 3.3 (1.0) | 3.0 (1.0)
  Intensity of services: OT Baseline | 2.0 (0.8) | 2.2 (0.9) | 2.3 (0.9) | 2.6 (0.8) | 2.6 (1.0)
  Intensity of services: OT 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Intensity of services: OT 6M | 2.1 (0.9) | 2.5 (1.0) | 2.6 (1.1) | 2.8 (1.0) | 2.8 (1.1)
  Intensity of services: OT 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Intensity of services: OT 12M | 2.0 (1.0) | 2.2 (1.0) | 2.5 (1.1) | 2.6 (0.9) | 2.5 (1.1)
  Intensity of services: OT 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Intensity of services: OT 18M | 2.1 (1.1) | 2.4 (1.0) | 2.5 (1.1) | 2.9 (1.0) | 2.6 (1.1)
  Intensity of services: OT 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Intensity of services: OT 24M | 2.0 (1.0) | 2.3 (1.1) | 2.4 (1.1) | 2.9 (1.0) | 2.5 (1.1)
  Intensity of services: ST: baseline | 1.7 (0.9) | 1.9 (1.0) | 2.0 (1.0) | 2.3 (1.0) | 2.4 (1.1)
  Intensity of services: ST: 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Intensity of services: ST: 6M | 1.8 (1.0) | 2.2 (1.2) | 2.1 (1.2) | 2.6 (1.2) | 2.6 (1.1)
  Intensity of services: ST: 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Intensity of services: ST: 12M | 1.7 (1.0) | 2.0 (1.2) | 1.9 (1.1) | 2.5 (1.1) | 2.4 (1.1)
  Intensity of services: ST: 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Intensity of services: ST: 18M | 1.8 (1.1) | 2.1 (1.2) | 2.2 (1.3) | 2.5 (1.2) | 2.7 (1.2)
  Intensity of services: ST: 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Intensity of services: ST: 24M | 1.7 (1.1) | 2.0 (1.2) | 2.0 (1.1) | 2.6 (1.3) | 2.5 (1.2)
  Family centeredness: Baseline | 3.5 (0.9) | 3.5 (0.8) | 3.5 (0.7) | 3.6 (0.7) | 3.5 (0.8)
  Family centeredness: 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Family centeredness: 6M | 3.4 (0.9) | 3.3 (0.9) | 3.5 (0.7) | 3.5 (0.8) | 3.4 (0.9)
  Family centeredness: 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Family centeredness: 12M | 3.4 (0.9) | 3.4 (0.9) | 3.4 (0.8) | 3.5 (0.8) | 3.4 (0.8)
  Family centeredness: 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Family centeredness: 18M | 3.2 (0.9) | 3.2 (0.9) | 3.3 (0.8) | 3.4 (0.9) | 3.2 (0.8)
  Family centeredness: 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Family centeredness: 24M | 3.2 (0.9) | 3.3 (0.9) | 3.3 (0.9) | 3.4 (0.9) | 3.3 (0.9)
  Services meeting needs AVG: Baseline | 3.7 (0.8) | 3.7 (0.8) | 3.5 (0.7) | 3.4 (0.7) | 3.3 (0.8)
  Services meeting needs AVG: 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Services meeting needs AVG: 6M | 3.8 (0.9) | 3.7 (0.8) | 3.5 (0.8) | 3.5 (0.8) | 3.3 (0.7)
  Services meeting needs AVG: 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Services meeting needs AVG: 12M | 3.8 (1.0) | 3.6 (0.8) | 3.5 (0.8) | 3.5 (0.7) | 3.3 (0.8)
  Services meeting needs AVG: 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Services meeting needs AVG: 18M | 3.7 (1.0) | 3.5 (0.9) | 3.4 (0.8) | 3.4 (0.8) | 3.1 (0.8)
  Services meeting needs AVG: 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Services meeting needs AVG: 24M | 3.8 (0.9) | 3.5 (0.9) | 3.5 (0.8) | 3.4 (0.8) | 3.1 (0.8)
  Focus of therapy, stretching muscles: Baseline | 3.8 (1.2) | 4.0 (1.2) | 4.0 (1.1) | 4.0 (1.1) | 4.1 (1.0)
  Focus of therapy, stretching muscles: 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Focus of therapy, stretching muscles: 6M | 3.7 (1.3) | 4.0 (1.2) | 4.1 (1.0) | 3.9 (1.2) | 4.1 (1.2)
  Focus of therapy, stretching muscles: 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Focus of therapy, stretching muscles: 12M | 3.8 (1.3) | 4.0 (1.1) | 4.0 (1.1) | 4.0 (1.1) | 3.9 (1.3)
  Focus of therapy, stretching muscles: 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Focus of therapy, stretching muscles: 18M | 3.7 (1.4) | 4.1 (1.1) | 4.0 (1.2) | 4.0 (1.1) | 4.0 (1.1)
  Focus of therapy, stretching muscles: 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Focus of therapy, stretching muscles: 24M | 3.8 (1.3) | 4.0 (1.2) | 3.9 (1.1) | 4.0 (1.1) | 3.9 (1.2)
  Focus of therapy, activities to improve: Baseline | 3.5 (1.5) | 4.0 (1.2) | 4.2 (1.0) | 3.9 (1.1) | 3.5 (1.3)
  Focus of therapy, activities to improve: 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Focus of therapy, activities to improve: 6M | 3.6 (1.4) | 3.8 (1.4) | 4.2 (1.0) | 3.9 (1.2) | 3.4 (1.5)
  Focus of therapy, activities to improve: 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Focus of therapy, activities to improve: 12M | 3.4 (1.5) | 3.8 (1.4) | 4.2 (1.0) | 4.0 (1.0) | 3.3 (1.4)
  Focus of therapy, activities to improve: 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Focus of therapy, activities to improve: 18M | 3.5 (1.5) | 3.9 (1.2) | 4.0 (1.2) | 3.9 (1.1) | 3.1 (1.4)
  Focus of therapy, activities to improve: 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Focus of therapy, activities to improve: 24M | 3.5 (1.5) | 3.7 (1.4) | 4.0 (1.1) | 3.8 (1.2) | 3.2 (1.4)
  Focus of therapy, health/well-being: Baseline | 3.0 (1.4) | 3.2 (1.3) | 3.1 (1.2) | 3.2 (1.3) | 2.9 (1.3)
  Focus of therapy, health/well-being: 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Focus of therapy, health/well-being: 6M | 3.1 (1.5) | 3.1 (1.4) | 3.1 (1.4) | 3.0 (1.3) | 3.0 (1.5)
  Focus of therapy, health/well-being: 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Focus of therapy, health/well-being: 12M | 2.9 (1.4) | 3.0 (1.4) | 3.1 (1.3) | 3.1 (1.3) | 2.8 (1.3)
  Focus of therapy, health/well-being: 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Focus of therapy, health/well-being: 18M | 2.8 (1.5) | 3.0 (1.4) | 2.9 (1.3) | 3.1 (1.3) | 2.6 (1.4)
  Focus of therapy, health/well-being: 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Focus of therapy, health/well-being: 24M | 2.9 (1.5) | 3.0 (1.5) | 2.9 (1.3) | 2.9 (1.4) | 2.7 (1.4)
  Focus of therapy, self-awareness: Baseline | 3.2 (1.4) | 3.1 (1.3) | 3.3 (1.2) | 3.3 (1.2) | 2.9 (1.4)
  Focus of therapy, self-awareness: 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Focus of therapy, self-awareness: 6M | 3.3 (1.4) | 3.1 (1.3) | 3.3 (1.3) | 3.3 (1.2) | 3.0 (1.4)
  Focus of therapy, self-awareness: 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Focus of therapy, self-awareness: 12M | 3.0 (1.4) | 3.3 (1.4) | 3.3 (1.3) | 3.2 (1.3) | 2.8 (1.4)
  Focus of therapy, self-awareness: 18M: number analyzed (Participants) | 148 | 101 | 48 | 83 | 75
  Focus of therapy, self-awareness: 18M | 3.2 (1.5) | 3.2 (1.4) | 3.0 (1.3) | 3.2 (1.4) | 2.6 (1.3)
  Focus of therapy, self-awareness: 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Focus of therapy, self-awareness: 24M | 3.1 (1.5) | 3.2 (1.5) | 3.4 (1.3) | 3.1 (1.3) | 2.7 (1.4)
  Focus of therapy, relaxation: Baseline | 3.3 (1.4) | 3.5 (1.3) | 3.8 (1.1) | 4.0 (1.1) | 4.0 (1.1)
  Focus of therapy, relaxation: 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Focus of therapy, relaxation: 6M | 3.4 (1.5) | 3.7 (1.2) | 4.1 (1.0) | 3.9 (1.1) | 4.1 (1.1)
  Focus of therapy, relaxation: 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Focus of therapy, relaxation: 12M | 3.3 (1.4) | 3.7 (1.3) | 3.7 (1.2) | 3.8 (1.2) | 3.9 (1.1)
  Focus of therapy, relaxation: 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Focus of therapy, relaxation: 18M | 3.4 (1.4) | 3.7 (1.3) | 3.6 (1.4) | 3.9 (1.1) | 3.9 (1.1)
  Focus of therapy, relaxation: 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Focus of therapy, relaxation: 24M | 3.3 (1.5) | 3.5 (1.4) | 3.5 (1.1) | 3.8 (1.2) | 3.8 (1.2)
  Focus of therapy, self-care routines: Baseline | 2.1 (1.3) | 2.4 (1.3) | 2.7 (1.2) | 2.5 (1.2) | 2.1 (1.4)
  Focus of therapy, self-care routines: 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Focus of therapy, self-care routines: 6M | 2.4 (1.4) | 2.7 (1.5) | 2.6 (1.3) | 2.5 (1.1) | 2.0 (1.3)
  Focus of therapy, self-care routines: 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Focus of therapy, self-care routines: 12M | 2.2 (1.3) | 2.6 (1.4) | 2.9 (1.3) | 2.4 (1.2) | 2.1 (1.2)
  Focus of therapy, self-care routines: 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Focus of therapy, self-care routines: 18M | 2.5 (1.5) | 2.5 (1.4) | 2.6 (1.4) | 2.4 (1.2) | 1.8 (1.1)
  Focus of therapy, self-care routines: 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Focus of therapy, self-care routines: 24M | 2.3 (1.4) | 2.3 (1.4) | 2.7 (1.3) | 2.5 (1.2) | 2.0 (1.2)
  Focus of therapy, assistive devices: Baseline | 2.6 (1.5) | 3.1 (1.4) | 3.6 (1.1) | 3.8 (1.1) | 3.7 (1.1)
  Focus of therapy, assistive devices: 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Focus of therapy, assistive devices: 6M | 2.6 (1.6) | 3.1 (1.5) | 3.3 (1.3) | 3.7 (1.2) | 3.8 (1.2)
  Focus of therapy, assistive devices: 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Focus of therapy, assistive devices: 12M | 2.4 (1.5) | 3.5 (1.4) | 3.6 (1.2) | 3.8 (1.1) | 3.5 (1.3)
  Focus of therapy, assistive devices: 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Focus of therapy, assistive devices: 18M | 2.7 (1.6) | 3.3 (1.5) | 3.4 (1.5) | 3.7 (1.2) | 3.5 (1.3)
  Focus of therapy, assistive devices: 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Focus of therapy, assistive devices: 24M | 2.4 (1.5) | 2.8 (1.6) | 3.4 (1.3) | 3.6 (1.2) | 3.6 (1.3)
  Focus of therapy, structured play: Baseline | 3.0 (1.5) | 3.2 (1.3) | 3.5 (1.2) | 3.4 (1.2) | 3.2 (1.2)
  Focus of therapy, structured play: 6M: number analyzed (Participants) | 148 | 105 | 49 | 84 | 85
  Focus of therapy, structured play: 6M | 3.1 (1.5) | 3.4 (1.3) | 3.6 (1.2) | 3.4 (1.2) | 3.2 (1.2)
  Focus of therapy, structured play: 12M: number analyzed (Participants) | 217 | 147 | 73 | 116 | 103
  Focus of therapy, structured play: 12M | 2.7 (1.5) | 3.1 (1.5) | 3.3 (1.2) | 3.3 (1.1) | 3.1 (1.2)
  Focus of therapy, structured play: 18M: number analyzed (Participants) | 147 | 101 | 48 | 83 | 75
  Focus of therapy, structured play: 18M | 3.0 (1.5) | 3.1 (1.4) | 3.2 (1.4) | 3.4 (1.1) | 3.0 (1.2)
  Focus of therapy, structured play: 24M: number analyzed (Participants) | 135 | 97 | 48 | 75 | 69
  Focus of therapy, structured play: 24M | 2.8 (1.5) | 2.8 (1.5) | 3.0 (1.4) | 3.1 (1.2) | 2.9 (1.2)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Participation outcome for the predictor family-centred service; Test type: Other; Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.06 to 2.02] — Data from all GMFCS levels was used, country was included as a model covariate. OR represents the odds of children developing 'better than expected' (top 10%) vs 'as expected' (central 80%) for each unit change in family-centredness outcome
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Participation outcome for the predictor parents' perception of needs being met; Test type: Other; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.07 to 2.03] — Country was included as a model covariate. OR represents the odds of children developing 'better than expected' (top 10%) vs 'as expected' (central 80%) for each unit change in parents' perception of needs being met
Statistical Analysis 3: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Participation outcome for the predictor degree of focus on environment (assistive devices, equipment, home/school modifications); Test type: Other; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.96 to 1.38] — Country was included as a model covariate. OR represents the odds of children developing 'better than expected' (top 10%) vs 'as expected' (central 80%) for each unit change in the amount of focus on environment
Statistical Analysis 4: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Participation outcome for the predictor focus on participation (structured play/recreation/leisure activities); Test type: Other; Odds Ratio (OR) = 1.30, 95% CI 2-sided [1.07 to 1.58] — Country was included as a model covariate. OR represents the odds of children developing 'better than expected' (top 10%) vs 'as expected' (central 80%) for each unit change in focus on participation
Statistical Analysis 5: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Participation outcome for the predictor amount of physical therapy services; Test type: Other; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.72 to 1.58] — Country was included as a model covariate. OR represents the odds of children developing 'better than expected' (top 10%) vs 'as expected' (central 80%) for each unit change in amount of physical therapy services
Statistical Analysis 6: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Participation outcome for the predictor amount of occupational therapy; Test type: Other; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.74 to 1.28] — Country was included as a model covariate. OR represents the odds of children developing 'better than expected' (top 10%) vs 'as expected' (central 80%) for each unit change in amount of occupational therapy services
Statistical Analysis 7: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Participation outcome for the predictor amount of speech and language therapy; Test type: Other; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.97 to 1.60] — Country was included as a model covariate. OR represents the odds of children developing 'better than expected' (top 10%) vs 'as expected' (central 80%) for each unit change in amount of speech and language therapy
Statistical Analysis 8: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Self Care outcome for the predictor family-centred service; Test type: Other; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.00 to 1.88] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 9: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Early Clinical Assessment of Balance outcome for the predictor family-centred service; Test type: Other; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.78 to 1.44] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 10: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Six Minute Walk Test outcome for the predictor family-centred service; Test type: Other; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.54 to 1.26] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 11: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Self Care outcome for the predictor parents' perception of needs being met; Test type: Other; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.00 to 1.87] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 12: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Early Clinical Assessment of Balance outcome for the predictor parents' perception of needs being met; Test type: Other; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.83 to 1.53] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 13: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Six Minute Walk Test outcome for the predictor parents' perception of needs being met; Test type: Other; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.59 to 1.3] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 14: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Self Care outcome for the predictor degree of focus on environment (assistive devices, equipment, home/school modifications); Test type: Other; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.9 to 1.29] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 15: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Early Clinical Assessment of Balance outcome for the predictor degree of focus on environment (assistive devices, equipment, home/school modifications); Test type: Other; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.86 to 1.22]
Statistical Analysis 16: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Six Minute Walk Test outcome for the predictor degree of focus on environment (assistive devices, equipment, home/school modifications); Test type: Other; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.7 to 1.13] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 17: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Self Care outcome for the predictor focus on participation (structured play/recreation/leisure activities); Test type: Other; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.9 to 1.31] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 18: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Early Clinical Assessment of Balance outcome for the predictor focus on participation (structured play/recreation/leisure activities); Test type: Other; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.91 to 1.32] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 19: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Six Minute Walk Test outcome for the predictor focus on participation (structured play/recreation/leisure activities); Test type: Other; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.76 to 1.24] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 20: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Self Care outcome for the predictor amount of physical therapy services; Test type: Other; Odds Ratio (OR) = 0.9, 95% CI 2-sided [.7 to 1.15] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 21: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Six Minute Walk Test outcome for the predictor amount of physical therapy services; Test type: Other; Odds Ratio (OR) = 1.05, 95% CI 2-sided [.74 to 1.48] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 22: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life -Self Care outcome for the predictor amount of occupational therapy; Test type: Other; Odds Ratio (OR) = .93, 95% CI 2-sided [.72 to 1.21] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 23: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Early Clinical Assessment of Balance outcome for the predictor amount of occupational therapy; Test type: Other; Odds Ratio (OR) = 1.15, 95% CI 2-sided [.89 to 1.5] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 24: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Six Minute Walk Test outcome for the predictor amount of occupational therapy; Test type: Other; Odds Ratio (OR) = .95, 95% CI 2-sided [.65 to 1.38] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 25: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Child Engagement in Daily Life - Self Care outcome for the predictor amount of speech and language therapy; Test type: Other; Odds Ratio (OR) = 1.03, 95% CI 2-sided [.81 to 1.31] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 26: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Early Clinical Assessment of Balance outcome for the predictor amount of speech and language therapy; Test type: Other; Odds Ratio (OR) = 1.1, 95% CI 2-sided [.87 to 1.39] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 27: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Six Minute Walk Test outcome for the predictor amount of speech and language therapy; Test type: Other; Odds Ratio (OR) = .86, 95% CI 2-sided [.6 to 1.25] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 28: Comparison: Gross Motor Function Classification System (GMFCS) Level I vs Gross Motor Function Classification System (GMFCS) Level II vs Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; Logistic regression comparing children progressing better than expected to those progressing as expected on the Early Clinical Assessment of Balance outcome for the predictor amount of physical therapy services; Test type: Other; Odds Ratio (OR) = 1.19, 95% CI 2-sided [.92 to 1.53] — [estimate comment as in outcome 9, analysis 2]

10. Secondary Outcome: Percentage of All Participants According to Gross Motor Function Classification System (GMFCS)
Description: The GMFCS is classification system based on functional body movement ability. GMFCS levels vary from I to V, with a level closest to I reflecting higher function. The general descriptions of a child at 6 to 12 years of age are: I: Walks without limitations; II: Walks with limitations; III: Walks using a hand-held mobility device; IV: Self-mobility with limitations; may use powered mobility; and V: Transported in manual wheelchair. Descriptors for the five levels vary by age of the child. Children were classified by consensus between parents and assessing therapists by comparing the child's functional movement ability to descriptors for each level of classification.
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Groups:
- Gross Motor Function Classification System (GMFCS) Level I: Participants scored on the GMFCS
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I
Number analyzed (Participants) | 708
percentage of participants
  GMFCS Level I | 32.1
  GMFCS Level II | 22.7
  GMFCS Level III | 11.3
  GMFCS Level IV | 18.2
  GMFCS Level V | 15.7

11. Secondary Outcome: Manual Ability Classification System (MACS)
Description: The MACS is a classification system based on functional hand movement ability. MACS levels vary from I to V, with a level closest to I reflecting higher function. The general descriptions for each level are: I: Handles objects easily & effectively; II: Handles most objects with somewhat reduced quality and/or speed; III: Handles objects with difficulty, needs help to prepare and/or modify activities; IV: Handles a limited selection of easily managed objects; and V: Does not handle objects and has severely limited ability to perform even simple actions.
Time Frame: Baseline consensus classification used for children 2 years and over at Baseline and 12M consensus classification used for children under 2 years at Baseline)
Population: Baseline consensus classification used for children 2 years and over at Baseline and 12M consensus classification used for children under 2 years at Baseline)
Measure: Number; unit: participants
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 227 | 161 | 80 | 129 | 111
participants
  MACS Level I | 95 | 33 | 12 | 4 | 0
  MACS Level II | 121 | 96 | 40 | 21 | 2
  MACS Level III | 9 | 24 | 21 | 49 | 4
  MACS Level IV | 2 | 8 | 6 | 49 | 52
  MACS Level V | 0 | 0 | 1 | 6 | 53

12. Secondary Outcome: Communication Function Classification System (CFCS)
Description: The CFCS is a classification system based on functional communication ability. CFCS levels vary from I to V, with a level closest to I reflecting higher function. The general descriptions for each level are: I: Effective sender/receiver with familiar/unfamiliar partners; II: Effective but slower paced sender and/or receiver with familiar/unfamiliar partners; III: Effective sender & receiver with familiar partners; IV: Inconsistent sender and/or receiver with familiar partners; and V: Seldom effective sender & receiver with familiar partners.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 227 | 161 | 80 | 129 | 111
participants
  CFCS Level I | 144 | 63 | 34 | 20 | 3
  CFCS Level II | 46 | 46 | 17 | 16 | 1
  CFCS Level III | 26 | 28 | 18 | 38 | 24
  CFCS Level IV | 10 | 23 | 9 | 45 | 42
  CFCS Level V | 1 | 1 | 2 | 10 | 41

13. Other Pre Specified Outcome: Physical Activity Measurement: StepWatch: Average Number of Strides Per Day Faster Than 30 Per Minute (Moderate- to High-intensity Strides)
Description: For participants who were ambulatory (GMFCS levels I, II, III), walking activity performance was measured within the context of daily life with a monitor called the StepWatch. It is a small (70 x 50 x 20 mm; 38 g), waterproof, self-contained device that is worn on the left ankle. Participants wore the StepWatch on their ankle (inside a knit cuff) each day for a seven-day sample. Specific variables reported are an intensity measure, average number of strides per day faster than 30 per minute (moderate to high intensity strides) for the seven-day sample.
Time Frame: up to 24-months
Population: StepWatch data was collected on a subset of 50 children in GMFCS Level I, II or II who participated in the Physical Activity Measurement Sub-Study. Children did not necessarily start the sub-study at the Baseline visit. Within each time point, there are two rows for age (under 6 years, 6 years and older).
Measure: Mean (Standard Deviation); unit: Strides per day faster than 30 /minute
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III
Number analyzed (Participants) | 23 | 20 | 7
Strides per day faster than 30 /minute
  StepWatch AVG strides/day >30/min: baseline <6yrs: number analyzed (Participants) | 1 | 3 | 1
  StepWatch AVG strides/day >30/min: baseline <6yrs | 1523.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 1185.0 (401.1) | 42.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  StepWatch AVG strides/day >30/min: baseline 6yrs +: number analyzed (Participants) | 5 | 7 | 2
  StepWatch AVG strides/day >30/min: baseline 6yrs + | 2930.2 (306.6) | 1691.3 (489.1) | 525.0 (125.8)
  StepWatch AVG strides/day >30/min: 6M <6yrs: number analyzed (Participants) | 5 | 4 | 1
  StepWatch AVG strides/day >30/min: 6M <6yrs | 1870.6 (907.3) | 1641.5 (711.8) | 0.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  StepWatch AVG strides/day >30/min: 6M 6yrs +: number analyzed (Participants) | 12 | 6 | 3
  StepWatch AVG strides/day >30/min: 6M 6yrs + | 2242.6 (1683.2) | 1892.9 (827.5) | 947.5 (481.1)
  StepWatch AVG strides/day >30/min: 12M <6yrs: number analyzed (Participants) | 4 | 4 | 2
  StepWatch AVG strides/day >30/min: 12M <6yrs | 2674.9 (1403.5) | 1262.0 (425.0) | 249.0 (321.0)
  StepWatch AVG strides/day >30/min: 12M 6yrs +: number analyzed (Participants) | 17 | 14 | 5
  StepWatch AVG strides/day >30/min: 12M 6yrs + | 2080.6 (923.7) | 1650.6 (801.6) | 721.1 (515.4)
  StepWatch AVG strides/day >30/min: 18M <6yrs: number analyzed (Participants) | 3 | 2 | 1
  StepWatch AVG strides/day >30/min: 18M <6yrs | 3530.3 (1128.6) | 1084.1 (593.8) | 673.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  StepWatch AVG strides/day >30/min: 18M 6yrs +: number analyzed (Participants) | 17 | 14 | 5
  StepWatch AVG strides/day >30/min: 18M 6yrs + | 2297.6 (822.7) | 1662.2 (725.0) | 429.9 (411.6)
  StepWatch AVG strides/day >30/min: 24M <6yrs: number analyzed (Participants) | 1 | 1 | 1
  StepWatch AVG strides/day >30/min: 24M <6yrs | 3066.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 653.9 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 1706.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  StepWatch AVG strides/day >30/min: 24M 6yrs +: number analyzed (Participants) | 15 | 16 | 4
  StepWatch AVG strides/day >30/min: 24M 6yrs + | 2766.8 (1054.7) | 1722.3 (862.6) | 587.4 (669.5)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; The outcome was modelled as a function of age using a linear mixed effects model, and the population value at age 12 years was estimated from the model; Test type: Other; population average = 2319, 95% CI 2-sided [1460 to 3218]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; [analysis description as in outcome 13, analysis 1]; Test type: Other; population average = 1858, 95% CI 2-sided [1233 to 2530]

14. Other Pre Specified Outcome: Physical Activity Measurement: StepWatch - Average Number of Single Leg Strides Per Day
Description: For participants who were ambulatory (GMFCS levels I, II, III), walking activity performance was measured within the context of daily life with a monitor called the StepWatch. It is a small (70 x 50 x 20 mm; 38 g), waterproof, self-contained device that is worn on the left ankle. Participants wore the StepWatch on their ankle (inside a knit cuff) each day for a seven-day sample. Specific variables reported are an an amount measure, average number of single leg strides per day for the seven-day sample.
Time Frame: up to 24-months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Avg number single leg strides per day
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III
Number analyzed (Participants) | 23 | 20 | 7
Avg number single leg strides per day
  StepWatch AVG SL strides/day: baseline <6yrs: number analyzed (Participants) | 1 | 3 | 1
  StepWatch AVG SL strides/day: baseline <6yrs | 4674.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 3622.7 (899.8) | 753.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  StepWatch AVG SL strides/day: baseline 6yrs +: number analyzed (Participants) | 5 | 7 | 2
  StepWatch AVG SL strides/day: baseline 6yrs + | 6548.2 (724.3) | 4196.7 (788.8) | 2173.3 (501.1)
  StepWatch AVG SL strides/day: 6M <6yrs: number analyzed (Participants) | 5 | 4 | 1
  StepWatch AVG SL strides/day: 6M <6yrs | 5031.7 (1720.0) | 3851.0 (751.8) | 140.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  StepWatch AVG SL strides/day: 6M 6yrs +: number analyzed (Participants) | 12 | 6 | 3
  StepWatch AVG SL strides/day: 6M 6yrs + | 5161.3 (2476.7) | 4733.5 (1445.4) | 2761.5 (851.5)
  StepWatch AVG SL strides/day: 12M <6yrs: number analyzed (Participants) | 4 | 4 | 2
  StepWatch AVG SL strides/day: 12M <6yrs | 6441.9 (2438.9) | 3669.1 (805.8) | 1829.5 (1883.0)
  StepWatch AVG SL strides/day: 12M 6yrs +: number analyzed (Participants) | 17 | 14 | 5
  StepWatch AVG SL strides/day: 12M 6yrs + | 5190.7 (1569.7) | 4329.3 (1550.3) | 2144.2 (1172.2)
  StepWatch AVG SL strides/day: 18M <6yrs: number analyzed (Participants) | 3 | 2 | 1
  StepWatch AVG SL strides/day: 18M <6yrs | 7205.3 (1387.3) | 3441.9 (1291.4) | 4083.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  StepWatch AVG SL strides/day: 18M 6yrs +: number analyzed (Participants) | 17 | 14 | 5
  StepWatch AVG SL strides/day: 18M 6yrs + | 5381.5 (1429.6) | 4116.6 (1023.0) | 1751.3 (1308.9)
  StepWatch AVG SL strides/day: 24M <6yrs: number analyzed (Participants) | 1 | 1 | 1
  StepWatch AVG SL strides/day: 24M <6yrs | 5956.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 2671.5 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 5559.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation
  StepWatch AVG SL strides/day: 24M 6yrs +: number analyzed (Participants) | 15 | 16 | 4
  StepWatch AVG SL strides/day: 24M 6yrs + | 6096.0 (1394.0) | 4014.7 (1507.4) | 1869.7 (1522.8)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; [analysis description as in outcome 13, analysis 1]; Test type: Other; population average = 5240, 95% CI 2-sided [3874 to 6670]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; [analysis description as in outcome 13, analysis 1]; Test type: Other; population average = 4319, 95% CI 2-sided [3258 to 5443]

15. Other Pre Specified Outcome: Physical Activity Measurement: Actigraph: Minutes of Moderate to Vigorous Physical Activity
Description: Participants wore a 3-dimensional accelerometer (Actigraph wGT3X) on their dominant wrist for a seven-day sample. Specific variables reported are number of minutes time spent in moderate/vigorous physical activity for a seven-day sample. The wrist mounted Actigraph counts were converted to waist worn activity counts.
Time Frame: up to 24-months
Population: Actigraph data was collected on a subset of 79 children who participated in the Physical Activity Measurement Sub-Study. Children did not necessarily start the sub-study at the Baseline visit. Within each time point, there are two rows for age (under 6 years, 6 years and older).
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 23 | 20 | 7 | 15 | 14
minutes per day
  Actigraph: min of Mod-Vig phys act, baseline <6yrs: number analyzed (Participants) | 1 | 3 | 1 | 3 | 2
  Actigraph: min of Mod-Vig phys act, baseline <6yrs | 230.3 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 98.7 (86.8) | 48.2 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 51.5 (24.2) | 76.2 (92.4)
  Actigraph: min of Mod-Vig phys act, baseline 6yrs+: number analyzed (Participants) | 5 | 7 | 2 | 6 | 4
  Actigraph: min of Mod-Vig phys act, baseline 6yrs+ | 190.9 (38.8) | 155.4 (52.8) | 26.2 (13.3) | 16.7 (23.1) | 8.8 (7.5)
  Actigraph: min of Mod-Vig phys act, 6M <6yrs: number analyzed (Participants) | 5 | 4 | 1 | 1 | 4
  Actigraph: min of Mod-Vig phys act, 6M <6yrs | 198.8 (63.6) | 122.1 (83.2) | 37.5 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 60.2 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 28.3 (54.8)
  Actigraph: min of Mod-Vig phys act, 6M 6yrs+: number analyzed (Participants) | 12 | 6 | 3 | 7 | 7
  Actigraph: min of Mod-Vig phys act, 6M 6yrs+ | 181.9 (50.9) | 126.3 (41.2) | 49.9 (17.5) | 15.8 (20.7) | 14.4 (14.1)
  Actigraph: min of Mod-Vig phys act, 12M <6yrs: number analyzed (Participants) | 4 | 4 | 2 | 3 | 4
  Actigraph: min of Mod-Vig phys act, 12M <6yrs | 222.8 (43.5) | 111.8 (64.7) | 56.4 (11.4) | 75.5 (34.1) | 38.7 (51.1)
  Actigraph: min of Mod-Vig phys act, 12M 6yrs+: number analyzed (Participants) | 17 | 14 | 5 | 11 | 8
  Actigraph: min of Mod-Vig phys act, 12M 6yrs+ | 156.4 (54.0) | 115.8 (39.4) | 26.3 (14.1) | 24.0 (27.9) | 19.4 (15.9)
  Actigraph: min of Mod-Vig phys act, 18M <6yrs: number analyzed (Participants) | 3 | 2 | 1 | 3 | 3
  Actigraph: min of Mod-Vig phys act, 18M <6yrs | 230.0 (17.2) | 56.2 (17.5) | 117.2 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 82.2 (68.5) | 49.5 (59.2)
  Actigraph: min of Mod-Vig phys act, 18M 6yrs+: number analyzed (Participants) | 17 | 14 | 5 | 11 | 10
  Actigraph: min of Mod-Vig phys act, 18M 6yrs+ | 166.2 (57.0) | 113.3 (51.9) | 32.6 (9.7) | 25.1 (31.1) | 14.9 (17.8)
  Actigraph: min of Mod-Vig phys act, 24M <6yrs: number analyzed (Participants) | 1 | 1 | 1 | 1 | 2
  Actigraph: min of Mod-Vig phys act, 24M <6yrs | 144.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 53.6 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 147.3 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 119.7 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 82.9 (28.4)
  Actigraph: min of Mod-Vig phys act, 24M 6yrs+: number analyzed (Participants) | 15 | 16 | 4 | 9 | 11
  Actigraph: min of Mod-Vig phys act, 24M 6yrs+ | 172.6 (40.6) | 105.9 (57.5) | 40.3 (18.5) | 34.5 (50.4) | 18.5 (30.7)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; [analysis description as in outcome 13, analysis 1]; Test type: Other; population average = 108, 95% CI 2-sided [67 to 151]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; [analysis description as in outcome 13, analysis 1]; Test type: Other; population average = 100, 95% CI 2-sided [58 to 145]
Statistical Analysis 3: Comparison: Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; The outcome was modelled as a function of age using a linear mixed effects model, and the population value at age 12 years was estimated from the model. This analysis combined children in GMFCS Levels III-V; Test type: Other; population average = 10, 95% CI 2-sided [0 to 35]

16. Other Pre Specified Outcome: Physical Activity Measurement: Actigraph: Average Physical Activity
Description: Participants wore a 3-dimensional accelerometer (Actigraph wGT3X) on their dominant wrist for a seven-day sample. Specific variables reported are average physical activity in raw activity counts per minute for a seven-day sample. The wrist mounted Actigraph counts were converted to waist worn activity counts.
Time Frame: up to 24-months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: counts per minute
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 23 | 20 | 7 | 15 | 14
counts per minute
  Actigraph: AVG phys act counts/min, baseline <6yrs: number analyzed (Participants) | 1 | 3 | 1 | 3 | 2
  Actigraph: AVG phys act counts/min, baseline <6yrs | 4642.6 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 3219.6 (1382.8) | 2560.7 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 2797.6 (694.2) | 3399.5 (2354.2)
  Actigraph: AVG phys act counts/min, baseline 6yrs: number analyzed (Participants) | 5 | 7 | 2 | 6 | 4
  Actigraph: AVG phys act counts/min, baseline 6yrs | 4655.4 (911.5) | 3556.4 (554.1) | 2012.7 (69.6) | 1567.4 (722.2) | 1321.4 (656.1)
  Actigraph: AVG phys act counts/min, 6M <6yrs: number analyzed (Participants) | 5 | 4 | 1 | 1 | 4
  Actigraph: AVG phys act counts/min, 6M <6yrs | 4519.4 (1032.4) | 3182.5 (1650.7) | 2785.6 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 2843.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 1687.6 (1271.4)
  Actigraph: AVG phys act counts/min, 6M 6yrs+: number analyzed (Participants) | 12 | 6 | 3 | 7 | 7
  Actigraph: AVG phys act counts/min, 6M 6yrs+ | 4258.2 (755.7) | 3502.8 (760.6) | 2524.7 (429.8) | 1775.5 (925.2) | 1737.0 (1080.6)
  Actigraph: AVG phys act counts/min, 12M <6yrs: number analyzed (Participants) | 4 | 4 | 2 | 3 | 4
  Actigraph: AVG phys act counts/min, 12M <6yrs | 4902.1 (805.3) | 3504.8 (932.7) | 2353.2 (511.0) | 3065.8 (1142.1) | 2810.5 (1276.7)
  Actigraph: AVG phys act counts/min, 12M 6yrs+: number analyzed (Participants) | 17 | 14 | 5 | 11 | 8
  Actigraph: AVG phys act counts/min, 12M 6yrs+ | 3587.2 (1349.9) | 3337.5 (742.7) | 2098.6 (563.1) | 1813.5 (826.4) | 1687.8 (752.5)
  Actigraph: AVG phys act counts/min, 18M <6yrs: number analyzed (Participants) | 3 | 2 | 1 | 3 | 3
  Actigraph: AVG phys act counts/min, 18M <6yrs | 5132.5 (512.3) | 2351.2 (236.0) | 4002.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 3217.0 (1320.1) | 2358.8 (1657.8)
  Actigraph: AVG phys act counts/min, 18M 6yrs+: number analyzed (Participants) | 17 | 14 | 5 | 11 | 10
  Actigraph: AVG phys act counts/min, 18M 6yrs+ | 4146.1 (1081.0) | 3280.7 (883.3) | 2286.8 (298.9) | 1835.5 (821.8) | 1561.2 (768.0)
  Actigraph: AVG phys act counts/min, 24M <6yrs: number analyzed (Participants) | 1 | 1 | 1 | 1 | 2
  Actigraph: AVG phys act counts/min, 24M <6yrs | 3454.9 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 2107.4 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 4211.5 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 4426.1 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 3292.2 (404.8)
  Actigraph: AVG phys act counts/min, 24M 6yrs+: number analyzed (Participants) | 15 | 16 | 4 | 9 | 11
  Actigraph: AVG phys act counts/min, 24M 6yrs+ | 4090.3 (678.8) | 3123.7 (866.2) | 2234.2 (616.3) | 1835.3 (934.8) | 1285.6 (639.9)
Statistical Analysis 1: Comparison: Gross Motor Function Classification System (GMFCS) Level I; [analysis description as in outcome 13, analysis 1]; Test type: Other; population average = 2815, 95% CI 2-sided [2025 to 3650]
Statistical Analysis 2: Comparison: Gross Motor Function Classification System (GMFCS) Level II; [analysis description as in outcome 13, analysis 1]; Test type: Other; population average = 3109, 95% CI 2-sided [2502 to 3739]
Statistical Analysis 3: Comparison: Gross Motor Function Classification System (GMFCS) Level III vs Gross Motor Function Classification System (GMFCS) Level IV vs Gross Motor Function Classification System (GMFCS) Level V; [analysis description as in outcome 15, analysis 3]; Test type: Other; population average = 1056, 95% CI 2-sided [471 to 1665]

17. Other Pre Specified Outcome: 1 Minute to 6 Minute Push Test (1MPT, 6MPT)
Description: The 1MPT to 6MPT are submaximal, clinical exercise tests, in which the total distance propelled in a manual wheelchair in 1-minute and 6-minutes, under controlled conditions, are measured for children who use a manual wheelchair for mobility (GMFCS level II, III, IV), the 1MPT/6MPT was conducted indoors or outdoors on a large, flat, hard terrain. A surveyor's measure wheel was used to calculate the total distance wheeled and a stopwatch to keep track of the allocated time. Standardized directions were used to encourage the child to wheel as far as possible. Distances wheeled (# of feet) are reported for a small number of participants within the Physical Activity sub-study.
Time Frame: up to 24-months
Population: The 1MPT and 6MPT were administered for exploratory purposes in the Physical Activity Measurement sub-study. The available N at each time point = 5 children or fewer. Not every child was tested at every time point.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 0 | 2 | 2 | 1 | 0
Feet
  1MPT, Baseline: under 6 years: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  1MPT, Baseline: under 6 years |  | 185.26 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 22.50 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 85.50 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |
  1MPT, Baseline: 6 years and older: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  1MPT, Baseline: 6 years and older |  | 232.20 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 86.00 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |  |
  1MPT, 6-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  1MPT, 6-month assessment: under 6 years |  |  | 45.60 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 89.10 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |
  1MPT, 6-month assessment: 6 years and older: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  1MPT, 6-month assessment: 6 years and older |  |  | 78.60 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |  |
  1MPT, 12-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  1MPT, 12-month assessment: under 6 years |  |  |  | 49.48 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |
  1MPT, 12-month assessment: 6 years and older: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  1MPT, 12-month assessment: 6 years and older |  |  | 101.85 (25.24) |  |
  1MPT, 18-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  1MPT, 18-month assessment: 6 years and older: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0
  1MPT, 18-month assessment: 6 years and older |  | 239.00 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 131.35 (44.05) |  |
  1MPT, 24-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  1MPT, 24-month assessment: 6 years and older: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0
  1MPT, 24-month assessment: 6 years and older |  |  | 95.60 (17.54) | 131.80 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |
  6MPT, Baseline: under 6 years: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  6MPT, Baseline: under 6 years |  | 1111.50 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 146.19 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 391.30 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |
  6MPT, Baseline: 6 years and older: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  6MPT, Baseline: 6 years and older |  | 1296.20 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 926.00 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |  |
  6MPT, 6-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  6MPT, 6-month assessment: under 6 years |  |  | 177.10 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 394.50 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |
  6MPT, 6-month assessment: 6 years and older: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  6MPT, 6-month assessment: 6 years and older |  |  | 435.50 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |  |
  6MPT, 12-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  6MPT, 12-month assessment: under 6 years |  |  |  | 296.89 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |
  6MPT, 12-month assessment: 6 years and older: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  6MPT, 12-month assessment: 6 years and older |  |  | 597.75 (71.77) |  |
  6MPT, 18-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  6MPT, 18-month assessment: 6 years and older: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0
  6MPT, 18-month assessment: 6 years and older |  | 1525.70 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 587.95 (133.57) |  |
  6MPT, 24-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  6MPT, 24-month assessment: 6 years and older: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0
  6MPT, 24-month assessment: 6 years and older |  |  | 422.85 (282.06) | 546.50 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |

18. Other Pre Specified Outcome: 1 Stroke Push Test (1SPT)
Description: The 1SPT is a clinical exercise test, in which the distance rolled in a manual wheelchair, under controlled conditions, with one push using both hands if possible is measured. Within this study a subsample of children who used a manual wheelchair for mobility (GMFCS levels III, IV) were tested on this measure. A surveyor's measure wheel will be used to calculate the total distance (# of feet) wheeled. Standardized directions are used to encourage the child to wheel as far as possible.
Time Frame: up to 24-months
Population: This test was administered for exploratory purposes in the Physical Activity Measurement sub-study. The available N at each time point is 4 or fewer. Also there are two age levels reported at each assessment time and children fell into only one of the two age groups.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 0 | 0 | 11 | 4 | 0
Feet
  1SPT, Baseline: under 6 years: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  1SPT, Baseline: under 6 years |  |  | 8.87 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 0.63 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |
  1SPT, Baseline: 6 years and older: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  1SPT, Baseline: 6 years and older |  |  | 5.73 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |  |
  1SPT 6-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  1SPT 6-month assessment: under 6 years |  |  | 10.87 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 1.40 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |
  1SPT 6-month assessment: 6 years and older: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  1SPT 6-month assessment: 6 years and older |  |  | 16.53 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |  |
  1SPT 12-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  1SPT 12-month assessment: under 6 years |  |  |  | 1.43 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |
  1SPT 12-month assessment: 6 years and older: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  1SPT 12-month assessment: 6 years and older |  |  | 6.30 (0.79) |  |
  1SPT 18-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  1SPT 18-month assessment: 6 years and older: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  1SPT 18-month assessment: 6 years and older |  |  | 10.29 (5.02) |  |
  1SPT 24-month assessment: under 6 years: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  1SPT 24-month assessment: 6 years and older: number analyzed (Participants) | 0 | 0 | 3 | 1 | 0
  1SPT 24-month assessment: 6 years and older |  |  | 12.01 (4.14) | 2.10 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation |

19. Other Pre Specified Outcome: Environment Section of the Participation and Environment Measure - Children and Youth (PEM-CY)
Description: The PEM-CY environment section is a caregiver completed 45-item questionnaire about the facilitators and barriers that might impact the child's participation in the home, school, and community environments. Twenty-five items include ratings on things that help or make it harder for the child to participate in activities in each environment (4-point scale from "not an issue" to "usually makes harder"). Twenty items include ratings of the availability of supports for the child's participation in each environment (4-point scale from "not needed" to "usually no"). Caregivers can also write in what family members do that help the child participate. A percentage score representing support for participation for each setting is calculated. The higher the percentage the more support the environment provides for the child's participation within the setting.
Time Frame: up to 24-months
Population: Caregiver PEM-CY data was collected on a subset of 79 children who participated in the Physical Activity Measurement Sub-Study. Children did not necessarily start the sub-study at the Baseline visit. Within each time point, there are two rows for age (under 6 years, 6 years and older).
Measure: Mean (Standard Deviation); unit: percentage of support for participation
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
Number analyzed (Participants) | 23 | 20 | 7 | 15 | 14
percentage of support for participation
  Support Participation HOME: baseline <6yrs: number analyzed (Participants) | 1 | 3 | 1 | 3 | 2
  Support Participation HOME: baseline <6yrs | 70 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 91.0 (8.5) | 85.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 69.6 (10.3) | 73.3 (9.4)
  Support Participation HOME: baseline 6yrs+: number analyzed (Participants) | 5 | 7 | 2 | 6 | 4
  Support Participation HOME: baseline 6yrs+ | 92.0 (7.4) | 78.0 (12.6) | 71.5 (9.2) | 81.7 (14.7) | 79.7 (9.6)
  Support Participation HOME: 6M <6yrs: number analyzed (Participants) | 5 | 4 | 1 | 1 | 4
  Support Participation HOME: 6M <6yrs | 93.2 (7.5) | 88.5 (1.0) | 88.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 70.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 77.8 (11.6)
  Support Participation HOME: 6M 6yrs+: number analyzed (Participants) | 12 | 6 | 3 | 7 | 7
  Support Participation HOME: 6M 6yrs+ | 93.6 (8.7) | 79.7 (7.3) | 80.0 (8.7) | 77.9 (11.4) | 78.4 (13.1)
  Support Participation HOME: 12M <6yrs: number analyzed (Participants) | 4 | 4 | 2 | 3 | 4
  Support Participation HOME: 12M <6yrs | 87.8 (14.3) | 93.5 (4.9) | 86.0 (8.5) | 73.7 (7.5) | 81.8 (17.1)
  Support Participation HOME: 12M 6yrs+: number analyzed (Participants) | 17 | 14 | 5 | 11 | 8
  Support Participation HOME: 12M 6yrs+ | 93.0 (9.1) | 84.0 (11.7) | 92.8 (4.8) | 79.0 (12.5) | 75.9 (11.2)
  Support Participation HOME: 18M <6yrs: number analyzed (Participants) | 3 | 2 | 1 | 3 | 3
  Support Participation HOME: 18M <6yrs | 87.7 (15.7) | 96.5 (2.1) | 90.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 92.0 (8.5) | 65.4 (16.7)
  Support Participation HOME: 18M 6yrs+: number analyzed (Participants) | 17 | 14 | 5 | 11 | 10
  Support Participation HOME: 18M 6yrs+ | 95.1 (9.1) | 87.3 (10.3) | 88.6 (10.9) | 71.8 (14.2) | 78.2 (10.2)
  Support Participation HOME: 24M <6yrs: number analyzed (Participants) | 1 | 1 | 1 | 1 | 2
  Support Participation HOME: 24M <6yrs | 86.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 85.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 83.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 75.6 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 68.2 (2.6)
  Support Participation HOME: 24M 6yrs+: number analyzed (Participants) | 15 | 16 | 4 | 9 | 11
  Support Participation HOME: 24M 6yrs+ | 93.8 (9.2) | 85.7 (10.4) | 80.8 (6.5) | 75.8 (12.7) | 75.6 (12.2)
  Support Participation COMMUNITY: baseline <6yrs: number analyzed (Participants) | 1 | 3 | 1 | 3 | 2
  Support Participation COMMUNITY: baseline <6yrs | 68.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 74.0 (20.4) | 85.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 61.2 (12.6) | 59.5 (3.5)
  Support Participation COMMUNITY: baseline 6yrs+: number analyzed (Participants) | 5 | 7 | 2 | 6 | 4
  Support Participation COMMUNITY: baseline 6yrs+ | 88.4 (13.6) | 70.9 (11.3) | 64.5 (3.5) | 65.2 (13.6) | 73.3 (7.8)
  Support Participation COMMUNITY: 6M <6yrs: number analyzed (Participants) | 5 | 4 | 1 | 1 | 4
  Support Participation COMMUNITY: 6M <6yrs | 81.6 (11.1) | 81.2 (8.3) | 85.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 48.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 69.8 (12.7)
  Support Participation COMMUNITY: 6M 6yrs+: number analyzed (Participants) | 12 | 6 | 3 | 7 | 7
  Support Participation COMMUNITY: 6M 6yrs+ | 90.4 (9.1) | 68.0 (15.3) | 62.0 (8.5) | 68.3 (14.6) | 74.6 (17.7)
  Support Participation COMMUNITY: 12M <6yrs: number analyzed (Participants) | 4 | 4 | 2 | 3 | 4
  Support Participation COMMUNITY: 12M <6yrs | 84.5 (12.0) | 86.0 (12.6) | 79.0 (1.4) | 61.0 (7.2) | 73.5 (16.0)
  Support Participation COMMUNITY: 12M 6yrs+: number analyzed (Participants) | 17 | 14 | 5 | 11 | 8
  Support Participation COMMUNITY: 12M 6yrs+ | 86.8 (11.4) | 72.4 (15.9) | 72.4 (14.7) | 66.7 (13.9) | 67.2 (16.1)
  Support Participation COMMUNITY: 18M <6yrs: number analyzed (Participants) | 3 | 2 | 1 | 3 | 3
  Support Participation COMMUNITY: 18M <6yrs | 91.7 (7.6) | 80.0 (0.0) | 75.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 60.0 (4.4) | 61.9 (13.7)
  Support Participation COMMUNITY: 18M 6yrs+: number analyzed (Participants) | 17 | 14 | 5 | 11 | 10
  Support Participation COMMUNITY: 18M 6yrs+ | 89.4 (10.8) | 73.9 (17.2) | 73.0 (9.1) | 65.7 (12.7) | 70.9 (12.1)
  Support Participation COMMUNITY: 24M <6yrs: number analyzed (Participants) | 1 | 1 | 1 | 1 | 2
  Support Participation COMMUNITY: 24M <6yrs | 87.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 83.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 75.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 59.9 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 59.1 (1.5)
  Support Participation COMMUNITY: 24M 6yrs+: number analyzed (Participants) | 15 | 16 | 4 | 9 | 11
  Support Participation COMMUNITY: 24M 6yrs+ | 90.0 (8.6) | 68.4 (23.8) | 67.5 (7.5) | 67.0 (13.7) | 66.4 (10.9)
  Support Participation SCHOOL: baseline <6yrs: number analyzed (Participants) | 1 | 3 | 1 | 3 | 2
  Support Participation SCHOOL: baseline <6yrs | 72.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 73.3 (26.3) | 80.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 66.9 (11.4) | 68.5 (0.7)
  Support Participation SCHOOL: baseline 6yrs+: number analyzed (Participants) | 5 | 7 | 2 | 6 | 4
  Support Participation SCHOOL: baseline 6yrs+ | 85.0 (8.0) | 76.6 (11.9) | 71.5 (2.1) | 76.7 (10.7) | 81.0 (10.8)
  Support Participation SCHOOL: 6M <6yrs: number analyzed (Participants) | 5 | 4 | 1 | 1 | 4
  Support Participation SCHOOL: 6M <6yrs | 83.8 (13.5) | 89.5 (4.2) | 86.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 73.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 70.0 (6.6)
  Support Participation SCHOOL: 6M 6yrs+: number analyzed (Participants) | 12 | 6 | 3 | 7 | 7
  Support Participation SCHOOL: 6M 6yrs+ | 87.4 (9.3) | 74.2 (11.9) | 72.3 (12.2) | 74.7 (15.1) | 81.5 (12.1)
  Support Participation SCHOOL: 12M <6yrs: number analyzed (Participants) | 4 | 4 | 2 | 3 | 4
  Support Participation SCHOOL: 12M <6yrs | 87.0 (12.4) | 93.0 (9.1) | 79.4 (6.5) | 70.0 (3.0) | 73.2 (11.9)
  Support Participation SCHOOL: 12M 6yrs+: number analyzed (Participants) | 17 | 14 | 5 | 11 | 8
  Support Participation SCHOOL: 12M 6yrs+ | 87.6 (10.8) | 75.5 (14.4) | 75.2 (9.2) | 75.0 (9.5) | 77.8 (12.7)
  Support Participation SCHOOL: 18M <6yrs: number analyzed (Participants) | 3 | 2 | 1 | 3 | 3
  Support Participation SCHOOL: 18M <6yrs | 94.3 (4.9) | 83.5 (0.7) | 70.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 76.3 (4.0) | 68.3 (5.6)
  Support Participation SCHOOL: 18M 6yrs+: number analyzed (Participants) | 17 | 14 | 5 | 11 | 10
  Support Participation SCHOOL: 18M 6yrs+ | 89.2 (7.9) | 77.2 (14.5) | 78.4 (13.5) | 71.6 (10.1) | 74.6 (11.0)
  Support Participation SCHOOL: 24M <6yrs: number analyzed (Participants) | 1 | 1 | 1 | 1 | 2
  Support Participation SCHOOL: 24M <6yrs | 80.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 91.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 75.0 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 69.1 (NA) — N/A when there is only 1 case in the cell therefore there is no standard deviation | 67.9 (1.3)
  Support Participation SCHOOL: 24M 6yrs+: number analyzed (Participants) | 15 | 16 | 4 | 9 | 11
  Support Participation SCHOOL: 24M 6yrs+ | 89.7 (10.2) | 78.0 (13.6) | 74.8 (12.5) | 71.9 (12.4) | 71.8 (7.4)

ADVERSE EVENTS:
Time Frame: 24 months
Description: Number of participant deaths during the course of involvement in the study. None of the deaths were study related.
Arm/Group | Gross Motor Function Classification System (GMFCS) Level I | Gross Motor Function Classification System (GMFCS) Level II | Gross Motor Function Classification System (GMFCS) Level III | Gross Motor Function Classification System (GMFCS) Level IV | Gross Motor Function Classification System (GMFCS) Level V
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/161 | 0/80 | 2/129 | 4/111
Serious Adverse Events (participants affected / at risk) | 0/227 | 0/161 | 0/80 | 0/129 | 0/111
Other Adverse Events (participants affected / at risk) | 0/227 | 0/161 | 0/80 | 0/129 | 0/111

LIMITATIONS AND CAVEATS:
This was a prospective observational cohort study not a randomized controlled trial. The Activity Performance sub-study included a smaller number of participants due to the extended week long data collection process.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No